CLINICAL TRIAL: NCT04047121
Title: Evaluation of Xeljanz Access Barriers Via Patient OOP Costs and TNFi Cycling
Brief Title: A Study to Evaluate Patient Characteristics and Treatment Patterns Among Rheumatoid Arthritis Patients
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A3921346
Record Dates: First submitted 2019-08-04; First posted 2019-08-06 (Actual); Results first posted 2020-10-19 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-06

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Truven Health MarketScan: The Truven Health MarketScan Research Databases reflects the combined healthcare service use of individuals covered by Truven Health clients (including employers, health plans, and hospitals) nationwide.

SUMMARY:
This is a retrospective cohort study to evaluate patient characteristics, treatment patterns including a 6-factor effectiveness proxy measure, health care resource use and associated costs among Rheumatoid Arthritis patients initiating treatment comparator groups of interest between January 2014 and September 2016 across three United States insurance claims databases.

ELIGIBILITY:
Inclusion Criteria:

* first pharmacy claim for Tofacitinib and then Etanercept or Adalimumab between Jan 2014 and Sep 2016 represents the index claim
* First, select patients receiving ≥1 Tofacitinib pharmacy claim (Jan 2014-Sep 2016) who did not have a Tofacitinib claim anytime prior to index
* Patients do have >1 advanced therapy filled on index date
* Physician diagnosis of Rheumatoid Arthritis (in any position) during the 1-year pre-index period, or on the index date
* Age 18+ years at index

Exclusion Criteria:

-None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients
Sampling Method: Probability Sample
Enrollment: 1349 (Actual)
Dates: Start 2019-05-20 (Actual); Primary Completion 2019-10-21 (Actual); Study Completion 2019-10-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, Collegeville, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A3921346

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 5-years data were retrieved from insurance claims Truven Health MarketScan Research Databases and were evaluated in 5 months of this retrospective, observational study. Participants who initiated treatment with tofacitinib, adalimumab or etanercept for rheumatoid arthritis (RA), between January 2014 and September 2016 were involved in this study.
Pre-assignment Details: 5-years (January 2012 to September 2017) included pre-index of 2 years, 2 years to capture treatment initiation (index date), and 1 year for follow-up post-index. Index date was first prescription date of treatment (tofacitinib, adalimumab or etanercept) from January 2014 to September 2016.
Groups:
- Tofacitinib Low Out of Pocket (OOP) Cost: Participants included in this reporting group were those who initiated tofacitinib between January 2014 and September 2016 and had low OOP cost (medical care expenses not reimbursed by insurance) as per data retrieved from insurance claims database.
- Tofacitinib High OOP Cost: Participants included in this reporting group were those who initiated tofacitinib between January 2014 and September 2016 and had high OOP cost (medical care expenses not reimbursed by insurance) as per data retrieved from insurance claims databases.
- Switch From Adalimumab to Etanercept: Participants included in this reporting group were those who initiated adalimumab between January 2014 and September 2016, and in this same duration switched from adalimumab to etanercept, as per data retrieved from insurance claims databases.
- Switch From Adalimumab to Tofacitinib: Participants included in this reporting group were those who initiated adalimumab between January 2014 and September 2016, and in this same duration switched from adalimumab to tofacitinib as per data retrieved from insurance claims databases.
- Switch From Etanercept to Adalimumab: Participants included in this reporting group were those who initiated etanercept between January 2014 and September 2016, and in this same duration switched from etanercept to adalimumab, as per data retrieved from insurance claims databases.
- Switch From Etanercept to Tofacitinib: Participants included in this reporting group were those who initiated etanercept between January 2014 and September 2016, and in this same duration switched from etanercept to tofacitinib, as per data retrieved from insurance claims databases.
Period: Overall Study
Arm/Group | Tofacitinib Low Out of Pocket (OOP) Cost | Tofacitinib High OOP Cost | Switch From Adalimumab to Etanercept | Switch From Adalimumab to Tofacitinib | Switch From Etanercept to Adalimumab | Switch From Etanercept to Tofacitinib
Started | 310 | 299 | 79 | 287 | 112 | 262
Completed | 310 | 299 | 79 | 287 | 112 | 262
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all eligible participants whose data were retrieved from databases and included in the study for retrospective observation.
Groups:
- Tofacitinib Low OOP Cost: Participants included in this reporting group were those who initiated tofacitinib between January 2014 and September 2016 and had low OOP cost (medical care expenses not reimbursed by insurance) as per data retrieved from insurance claims database.
- Total: Total of all reporting groups
Arm/Group | Tofacitinib Low OOP Cost | Tofacitinib High OOP Cost | Switch From Adalimumab to Etanercept | Switch From Adalimumab to Tofacitinib | Switch From Etanercept to Adalimumab | Switch From Etanercept to Tofacitinib | Total
Number analyzed (Participants) | 310 | 299 | 79 | 287 | 112 | 262 | 1349
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.67 (12.93) | 54.44 (11.01) | 50.52 (11.60) | 55.15 (11.14) | 53.36 (12.05) | 54.50 (12.25) | 55.26 (12.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 248 | 240 | 62 | 243 | 85 | 219 | 1097
  Male | 62 | 59 | 17 | 44 | 27 | 43 | 252
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Geographic Region [Count of Participants; unit: Participants]
  Northeast Region | 97 | 61 | 12 | 58 | 17 | 57 | 302
  North Central Region | 68 | 61 | 16 | 55 | 30 | 43 | 273
  South Region | 108 | 135 | 41 | 137 | 41 | 128 | 590
  West Region | 37 | 42 | 10 | 34 | 24 | 34 | 181
  Unknown Region | 0 | 0 | 0 | 3 | 0 | 0 | 3
Pre-index Biologic Disease Modifying Antirheumatic Drugs (bDMARDs) Use [Count of Participants; unit: Participants] — Participants who took bDMARDs before index date were reported.
  Participants | 0 | 0 | 52 | 238 | 87 | 224 | 601
Pre-index Non-biological Disease Modifying Antirheumatic Drug (NB-DMARDs) Use [Count of Participants; unit: Participants] — Participants who took NB-DMARDs before index date were reported.
  Participants | 245 | 243 | 64 | 226 | 79 | 198 | 1055
Disease Duration [Mean (Standard Deviation); unit: Days] — The number of days from the earliest claim with a diagnosis of RA within pre-index duration until the index date were identified and reported.
  Days | 511.92 (310.83) | 563.50 (317.53) | 452.04 (254.00) | 685.60 (313.28) | 432.03 (216.31) | 640.35 (278.94) | 575.11 (308.02)
Pre-index Claims-based Index For Rheumatoid Arthritis Severity (CIRAS) [Mean (Standard Deviation); unit: Units on a scale] — CIRAS provided a single value of rheumatoid arthritis severity using the following 9 measures: age, gender, inflammatory marker tests, rehabilitation visits, felty Syndrome, platelet orders, rheumatoid factor tests, chemistry panels, and rheumatologist visits. Type, or amount present, of all 9 measures was used to derive the overall CIRAS score by applying a weighted average. The CIRAS score was observed to range from 0-9.58 in this study, with higher values indicating generally greater severity of RA.
  Units on a scale | 4.50 (1.62) | 4.94 (1.48) | 5.15 (1.51) | 4.71 (1.44) | 4.61 (1.29) | 4.65 (1.47) | 4.72 (1.50)
Quan-Charlson Score [Count of Participants; unit: Participants] — The Quan-Charlson comorbidity index (QCCI) score predicts the probability of death in participants and was based on the presence of any International Classification of Diseases (ICD) diagnosis codes on medical claims at any time during pre-index period. Total score ranges from 0 to 9.0. A score of zero indicates that no comorbidities were found. The higher the score, the more likely the predicted outcome could result in mortality. Here, participants with QCCI score 0, 1 to 2, 3 to 4, and 5 or more were reported.
  Participants
    0 | 1 | 0 | 0 | 0 | 2 | 1 | 4
    1-2 | 235 | 244 | 65 | 226 | 91 | 208 | 1069
    3-4 | 52 | 46 | 10 | 52 | 15 | 37 | 212
    Greater than or equal to (>=) 5 | 22 | 9 | 4 | 9 | 4 | 16 | 64

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Were Persistent With Index Medication During 12 Months Post-index Date
Description: Persistent with the index medication was defined as not having a gap in the therapy of at least 60 days between prescription fill dates and their administration. Index medications were tofacitinib, adalimumab or etanercept.
Time Frame: During 12 months post-index date
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | Tofacitinib Low OOP Cost | Tofacitinib High OOP Cost | Switch From Adalimumab to Etanercept | Switch From Adalimumab to Tofacitinib | Switch From Etanercept to Adalimumab | Switch From Etanercept to Tofacitinib
Number analyzed (Participants) | 310 | 299 | 79 | 287 | 112 | 262
Percentage of participants | 47.42 | 42.81 | 36.71 | 50.52 | 38.39 | 45.80
Statistical Analysis 1: Comparison: Tofacitinib Low OOP Cost vs Tofacitinib High OOP Cost; Test type: Superiority; p = 0.2531, Chi-squared
Statistical Analysis 2: Comparison: Switch From Adalimumab to Etanercept vs Switch From Adalimumab to Tofacitinib; Test type: Superiority; p = 0.0295, Chi-squared
Statistical Analysis 3: Comparison: Switch From Etanercept to Adalimumab vs Switch From Etanercept to Tofacitinib; Test type: Superiority; p = 0.1857, Chi-squared
Statistical Analysis 4: Comparison: Tofacitinib Low OOP Cost vs Tofacitinib High OOP Cost; To control and remove the possible influence of the independent variables (like treatment cohort, demographic and clinical characteristics of interest, etc. and clinical judgement.) on the outcome measure, multivariable analysis was performed; Test type: Superiority; p = 0.3297, Regression, Logistic; Odds Ratio (OR) = 0.8401, 95% CI 2-sided [0.5919 to 1.1925]
Statistical Analysis 5: Comparison: Switch From Adalimumab to Etanercept vs Switch From Adalimumab to Tofacitinib; [analysis description as in outcome 1, analysis 4]; Test type: Superiority; p = 0.2003, Regression, Logistic; Odds Ratio (OR) = 1.5066, 95% CI 2-sided [0.8046 to 2.8209]
Statistical Analysis 6: Comparison: Switch From Etanercept to Adalimumab vs Switch From Etanercept to Tofacitinib; [analysis description as in outcome 1, analysis 4]; Test type: Superiority; p = 0.2276, Regression, Logistic; Odds Ratio (OR) = 1.4052, 95% CI 2-sided [0.8086 to 2.4420]

2. Primary Outcome: Percentage of Participants Who Immediately Switched Index Medication During 12 Months Post-index Date
Description: Participants who switched from index medication immediately were those who initiated a non-index advanced therapy before end of a 60-day gap in index medication. Index medications were tofacitinib, adalimumab or etanercept.
Time Frame: During 12 months post-index date
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | Tofacitinib Low OOP Cost | Tofacitinib High OOP Cost | Switch From Adalimumab to Etanercept | Switch From Adalimumab to Tofacitinib | Switch From Etanercept to Adalimumab | Switch From Etanercept to Tofacitinib
Number analyzed (Participants) | 310 | 299 | 79 | 287 | 112 | 262
Percentage of participants | 10.32 | 10.70 | 22.78 | 15.33 | 25.89 | 22.90
Statistical Analysis 1: Comparison: Tofacitinib Low OOP Cost vs Tofacitinib High OOP Cost; Test type: Superiority; p = 0.8786, Chi-squared
Statistical Analysis 2: Comparison: Switch From Adalimumab to Etanercept vs Switch From Adalimumab to Tofacitinib; Test type: Superiority; p = 0.1178, Chi-squared
Statistical Analysis 3: Comparison: Switch From Etanercept to Adalimumab vs Switch From Etanercept to Tofacitinib; Test type: Superiority; p = 0.5337, Chi-squared
Statistical Analysis 4: Comparison: Tofacitinib Low OOP Cost vs Tofacitinib High OOP Cost; [analysis description as in outcome 1, analysis 4]; Test type: Superiority; p = 0.9212, Regression, Logistic; Odds Ratio (OR) = 1.0283, 95% CI 2-sided [0.5911 to 1.7890]
Statistical Analysis 5: Comparison: Switch From Adalimumab to Etanercept vs Switch From Adalimumab to Tofacitinib; [analysis description as in outcome 1, analysis 4]; Test type: Superiority; p = 0.4693, Regression, Logistic; Odds Ratio (OR) = 0.7464, 95% CI 2-sided [0.3380 to 1.6482]
Statistical Analysis 6: Comparison: Switch From Etanercept to Adalimumab vs Switch From Etanercept to Tofacitinib; [analysis description as in outcome 1, analysis 4]; Test type: Superiority; p = 0.5593, Regression, Logistic; Odds Ratio (OR) = 0.8212, 95% CI 2-sided [0.4239 to 1.5910]

3. Primary Outcome: Percentage of Participants Who Discontinued Then Switched Index Medication During 12 Months Post-index Date
Description: Participants who discontinued index medication then switched from index medication were those who had gap in the index medication therapy of at least 60 days and then after the gap they switched to an advanced therapy different from index medication. Index medications were tofacitinib, adalimumab or etanercept.
Time Frame: During 12 months post-index date
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | Tofacitinib Low OOP Cost | Tofacitinib High OOP Cost | Switch From Adalimumab to Etanercept | Switch From Adalimumab to Tofacitinib | Switch From Etanercept to Adalimumab | Switch From Etanercept to Tofacitinib
Number analyzed (Participants) | 310 | 299 | 79 | 287 | 112 | 262
Percentage of participants | 3.87 | 4.68 | 8.86 | 6.62 | 7.14 | 5.34
Statistical Analysis 1: Comparison: Tofacitinib Low OOP Cost vs Tofacitinib High OOP Cost; Test type: Superiority; p = 0.6205, Chi-squared
Statistical Analysis 2: Comparison: Switch From Adalimumab to Etanercept vs Switch From Adalimumab to Tofacitinib; Test type: Superiority; p = 0.4924, Chi-squared
Statistical Analysis 3: Comparison: Switch From Etanercept to Adalimumab vs Switch From Etanercept to Tofacitinib; Test type: Superiority; p = 0.4982, Chi-squared
Statistical Analysis 4: Comparison: Tofacitinib Low OOP Cost vs Tofacitinib High OOP Cost; [analysis description as in outcome 1, analysis 4]; Test type: Superiority; p = 0.5494, Regression, Logistic; Odds Ratio (OR) = 1.3182, 95% CI 2-sided [0.5335 to 3.2570]
Statistical Analysis 5: Comparison: Switch From Etanercept to Adalimumab vs Switch From Etanercept to Tofacitinib; [analysis description as in outcome 1, analysis 4]; Test type: Superiority; p = 0.7830, Regression, Logistic; Odds Ratio (OR) = 1.1664, 95% CI 2-sided [0.3900 to 3.4883]

4. Primary Outcome: Percentage of Participants Who Discontinued Then Restarted Index Medication During 12 Months Post-index Date
Description: Participants who discontinued index medication and then restarted index medication were those who had a gap in the index medication therapy of at least 60 days and the first advanced therapy observed after the gap was the index medication. Index medications were tofacitinib, adalimumab or etanercept.
Time Frame: During 12 months post index date
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | Tofacitinib Low OOP Cost | Tofacitinib High OOP Cost | Switch From Adalimumab to Etanercept | Switch From Adalimumab to Tofacitinib | Switch From Etanercept to Adalimumab | Switch From Etanercept to Tofacitinib
Number analyzed (Participants) | 310 | 299 | 79 | 287 | 112 | 262
Percentage of participants | 13.23 | 15.72 | 11.39 | 10.10 | 11.61 | 10.69
Statistical Analysis 1: Comparison: Tofacitinib Low OOP Cost vs Tofacitinib High OOP Cost; Test type: Superiority; p = 0.3817, Chi-squared
Statistical Analysis 2: Comparison: Switch From Adalimumab to Etanercept vs Switch From Adalimumab to Tofacitinib; Test type: Superiority; p = 0.7397, Chi-squared
Statistical Analysis 3: Comparison: Switch From Etanercept to Adalimumab vs Switch From Etanercept to Tofacitinib; Test type: Superiority; p = 0.7942, Chi-squared
Statistical Analysis 4: Comparison: Tofacitinib Low OOP Cost vs Tofacitinib High OOP Cost; [analysis description as in outcome 1, analysis 4]; Test type: Superiority; p = 0.7924, Regression, Logistic; Odds Ratio (OR) = 1.0682, 95% CI 2-sided [0.6537 to 1.7455]
Statistical Analysis 5: Comparison: Switch From Adalimumab to Etanercept vs Switch From Adalimumab to Tofacitinib; [analysis description as in outcome 1, analysis 4]; Test type: Superiority; p = 0.9339, Regression, Logistic; Odds Ratio (OR) = 1.0414, 95% CI 2-sided [0.3997 to 2.7134]
Statistical Analysis 6: Comparison: Switch From Etanercept to Adalimumab vs Switch From Etanercept to Tofacitinib; [analysis description as in outcome 1, analysis 4]; Test type: Superiority; p = 0.6497, Regression, Logistic; Odds Ratio (OR) = 0.8195, 95% CI 2-sided [0.3470 to 1.9350]

5. Primary Outcome: Percentage of Participants Who Discontinued Without Switching or Restarting Index Medication During 12 Months Post-index Date
Description: Participants who discontinued index medication without switching or restarting index medication were those who had a gap in index medication therapy of at least 60 days and there were no claims for either the index medication or a different advanced therapy for the remainder of the follow-up period. Index medications were tofacitinib, adalimumab or etanercept.
Time Frame: During 12 months post index date
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | Tofacitinib Low OOP Cost | Tofacitinib High OOP Cost | Switch From Adalimumab to Etanercept | Switch From Adalimumab to Tofacitinib | Switch From Etanercept to Adalimumab | Switch From Etanercept to Tofacitinib
Number analyzed (Participants) | 310 | 299 | 79 | 287 | 112 | 262
Percentage of participants | 25.16 | 26.09 | 20.25 | 17.42 | 16.96 | 15.27
Statistical Analysis 1: Comparison: Tofacitinib Low OOP Cost vs Tofacitinib High OOP Cost; Test type: Superiority; p = 0.7936, Chi-squared
Statistical Analysis 2: Comparison: Switch From Adalimumab to Etanercept vs Switch From Adalimumab to Tofacitinib; Test type: Superiority; p = 0.5621, Chi-squared
Statistical Analysis 3: Comparison: Switch From Etanercept to Adalimumab vs Switch From Etanercept to Tofacitinib; Test type: Superiority; p = 0.6800, Chi-squared
Statistical Analysis 4: Comparison: Tofacitinib Low OOP Cost vs Tofacitinib High OOP Cost; [analysis description as in outcome 1, analysis 4]; Test type: Superiority; p = 0.5051, Regression, Logistic; Odds Ratio (OR) = 1.1438, 95% CI 2-sided [0.7705 to 1.6978]
Statistical Analysis 5: Comparison: Switch From Adalimumab to Etanercept vs Switch From Adalimumab to Tofacitinib; [analysis description as in outcome 1, analysis 4]; Test type: Superiority; p = 0.7131, Regression, Logistic; Odds Ratio (OR) = 0.8576, 95% CI 2-sided [0.3781 to 1.9452]
Statistical Analysis 6: Comparison: Switch From Etanercept to Adalimumab vs Switch From Etanercept to Tofacitinib; [analysis description as in outcome 1, analysis 4]; Test type: Superiority; p = 0.6490, Regression, Logistic; Odds Ratio (OR) = 0.8415, 95% CI 2-sided [0.4003 to 1.7690]

6. Secondary Outcome: Percentage of Participants Who Switched Index Medication Any Time During 12 Months Post-index Date
Description: Participants who switched from index medication at any time during the 12-month follow-up post-index period were evaluated. Index medications were tofacitinib, adalimumab or etanercept.
Time Frame: During 12 months post-index date
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | Tofacitinib Low OOP Cost | Tofacitinib High OOP Cost | Switch From Adalimumab to Etanercept | Switch From Adalimumab to Tofacitinib | Switch From Etanercept to Adalimumab | Switch From Etanercept to Tofacitinib
Number analyzed (Participants) | 310 | 299 | 79 | 287 | 112 | 262
Percentage of participants | 14.19 | 16.05 | 34.18 | 23.00 | 35.71 | 29.77
Statistical Analysis 1: Comparison: Tofacitinib Low OOP Cost vs Tofacitinib High OOP Cost; Test type: Superiority; p = 0.5217, Chi-squared
Statistical Analysis 2: Comparison: Switch From Adalimumab to Etanercept vs Switch From Adalimumab to Tofacitinib; Test type: Superiority; p = 0.0432, Chi-squared
Statistical Analysis 3: Comparison: Switch From Etanercept to Adalimumab vs Switch From Etanercept to Tofacitinib; Test type: Superiority; p = 0.2573, Chi-squared
Statistical Analysis 4: Comparison: Tofacitinib Low OOP Cost vs Tofacitinib High OOP Cost; [analysis description as in outcome 1, analysis 4]; Test type: Superiority; p = 0.5368, Regression, Logistic; Odds Ratio (OR) = 1.1637, 95% CI 2-sided [0.7193 to 1.8827]
Statistical Analysis 5: Comparison: Switch From Adalimumab to Etanercept vs Switch From Adalimumab to Tofacitinib; [analysis description as in outcome 1, analysis 4]; Test type: Superiority; p = 0.4685, Regression, Logistic; Odds Ratio (OR) = 0.7757, 95% CI 2-sided [0.3904 to 1.5413]
Statistical Analysis 6: Comparison: Switch From Etanercept to Adalimumab vs Switch From Etanercept to Tofacitinib; [analysis description as in outcome 1, analysis 4]; Test type: Superiority; p = 0.3112, Regression, Logistic; Odds Ratio (OR) = 0.7354, 95% CI 2-sided [0.4057 to 1.3330]

7. Secondary Outcome: Mean of Number of Days to Immediate Switch From Index Medication During 12 Months Post-index Date
Description: Participants who switched from index medication immediately were those who initiated a non-index advanced therapy before the end of a 60-day gap in index medication. Index medications were tofacitinib, adalimumab or etanercept. Number of days to immediately switch from index medication = immediate switch date - index date + 1.
Time Frame: During 12 months post-index date
Population: Analysis was performed on all eligible participants whose data were retrieved from databases and included in the study for retrospective observation. Here, "Overall Number of Participants Analyzed" refers to participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Tofacitinib Low OOP Cost | Tofacitinib High OOP Cost | Switch From Adalimumab to Etanercept | Switch From Adalimumab to Tofacitinib | Switch From Etanercept to Adalimumab | Switch From Etanercept to Tofacitinib
Number analyzed (Participants) | 32 | 32 | 18 | 44 | 29 | 60
Days | 155.00 (91.02) | 149.56 (88.40) | 144.00 (59.64) | 125.84 (84.73) | 148.69 (73.22) | 145.37 (87.59)
Statistical Analysis 1: Comparison: Tofacitinib Low OOP Cost vs Tofacitinib High OOP Cost; Test type: Superiority; p = 0.8122, Log Rank
Statistical Analysis 2: Comparison: Switch From Adalimumab to Etanercept vs Switch From Adalimumab to Tofacitinib; Test type: Superiority; p = 0.7766, Log Rank
Statistical Analysis 3: Comparison: Switch From Etanercept to Adalimumab vs Switch From Etanercept to Tofacitinib; Test type: Superiority; p = 0.8305, Log Rank
Statistical Analysis 4: Comparison: Tofacitinib Low OOP Cost vs Tofacitinib High OOP Cost; [analysis description as in outcome 1, analysis 4]; Test type: Superiority; p = 0.1845, Regression, Cox; Hazard Ratio (HR) = 0.5814, 95% CI 2-sided [0.2610 to 1.2952]
Statistical Analysis 5: Comparison: Switch From Adalimumab to Etanercept vs Switch From Adalimumab to Tofacitinib; [analysis description as in outcome 1, analysis 4]; Test type: Superiority; p = 0.2951, Regression, Cox; Hazard Ratio (HR) = 1.5908, 95% CI 2-sided [0.6671 to 3.7936]
Statistical Analysis 6: Comparison: Switch From Etanercept to Adalimumab vs Switch From Etanercept to Tofacitinib; [analysis description as in outcome 1, analysis 4]; Test type: Superiority; p = 0.4907, Regression, Cox; Hazard Ratio (HR) = 1.3546, 95% CI 2-sided [0.6584 to 2.7870]

8. Secondary Outcome: Mean of Number of Days to Immediate or Delayed Switch Index Medication During 12 Months Post-index Date
Description: Number of days to immediate or delayed switch from index medication any time during the 12-month follow-up period = immediate or delayed switch date - index date + 1. Index medications were tofacitinib, adalimumab or etanercept.
Time Frame: During 12 month post-index date
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Tofacitinib Low OOP Cost | Tofacitinib High OOP Cost | Switch From Adalimumab to Etanercept | Switch From Adalimumab to Tofacitinib | Switch From Etanercept to Adalimumab | Switch From Etanercept to Tofacitinib
Number analyzed (Participants) | 44 | 48 | 27 | 66 | 40 | 78
Days | 168.11 (84.29) | 175.98 (90.52) | 182.70 (83.90) | 158.71 (90.81) | 170.73 (81.64) | 169.36 (96.58)
Statistical Analysis 1: Comparison: Tofacitinib Low OOP Cost vs Tofacitinib High OOP Cost; Test type: Superiority; p = 0.6006, Log Rank
Statistical Analysis 2: Comparison: Switch From Adalimumab to Etanercept vs Switch From Adalimumab to Tofacitinib; Test type: Superiority; p = 0.2941, Log Rank
Statistical Analysis 3: Comparison: Switch From Etanercept to Adalimumab vs Switch From Etanercept to Tofacitinib; Test type: Superiority; p = 0.9610, Log Rank
Statistical Analysis 4: Comparison: Tofacitinib Low OOP Cost vs Tofacitinib High OOP Cost; [analysis description as in outcome 1, analysis 4]; Test type: Superiority; p = 0.0455, Regression, Cox; Hazard Ratio (HR) = 0.5571, 95% CI 2-sided [0.3140 to 0.9884]
Statistical Analysis 5: Comparison: Switch From Adalimumab to Etanercept vs Switch From Adalimumab to Tofacitinib; [analysis description as in outcome 1, analysis 4]; Test type: Superiority; p = 0.0274, Regression, Cox; Hazard Ratio (HR) = 2.1781, 95% CI 2-sided [1.0904 to 4.3506]
Statistical Analysis 6: Comparison: Switch From Etanercept to Adalimumab vs Switch From Etanercept to Tofacitinib; [analysis description as in outcome 1, analysis 4]; Test type: Superiority; p = 0.6787, Regression, Cox; Hazard Ratio (HR) = 0.8896, 95% CI 2-sided [0.5114 to 1.5475]

9. Secondary Outcome: Mean of Number of Days to Discontinue Index Medication During 12 Months Post-index Date
Description: Number of days to discontinue index medication = date of last persistent index medication prescription/administration + days supply- index date + 1. Index medications were tofacitinib, adalimumab or etanercept. Persistent with the index medication was defined as not having a gap in the therapy of at least 60 days between prescription fill dates and their administration.
Time Frame: During 12 months post-index date
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Tofacitinib Low OOP Cost | Tofacitinib High OOP Cost | Switch From Adalimumab to Etanercept | Switch From Adalimumab to Tofacitinib | Switch From Etanercept to Adalimumab | Switch From Etanercept to Tofacitinib
Number analyzed (Participants) | 158 | 168 | 50 | 139 | 68 | 138
Days | 119.62 (80.01) | 106.17 (76.50) | 111.74 (74.97) | 109.42 (74.16) | 130.18 (70.71) | 118.91 (77.58)
Statistical Analysis 1: Comparison: Tofacitinib Low OOP Cost vs Tofacitinib High OOP Cost; Test type: Superiority; p = 0.9084, Log Rank
Statistical Analysis 2: Comparison: Switch From Adalimumab to Etanercept vs Switch From Adalimumab to Tofacitinib; Test type: Superiority; p = 0.8325, Log Rank
Statistical Analysis 3: Comparison: Switch From Etanercept to Adalimumab vs Switch From Etanercept to Tofacitinib; Test type: Superiority; p = 0.9630, Log Rank
Statistical Analysis 4: Comparison: Tofacitinib Low OOP Cost vs Tofacitinib High OOP Cost; [analysis description as in outcome 1, analysis 4]; Test type: Superiority; p = 0.7909, Regression, Cox; Hazard Ratio (HR) = 1.0508, 95% CI 2-sided [0.7284 to 1.5160]
Statistical Analysis 5: Comparison: Switch From Adalimumab to Etanercept vs Switch From Adalimumab to Tofacitinib; [analysis description as in outcome 1, analysis 4]; Test type: Superiority; p = 0.6027, Regression, Cox; Hazard Ratio (HR) = 0.8117, 95% CI 2-sided [0.3700 to 1.7808]
Statistical Analysis 6: Comparison: Switch From Etanercept to Adalimumab vs Switch From Etanercept to Tofacitinib; [analysis description as in outcome 1, analysis 4]; Test type: Superiority; p = 0.6978, Regression, Cox; Hazard Ratio (HR) = 1.1742, 95% CI 2-sided [0.5222 to 2.6404]

10. Secondary Outcome: Duration of Index Medication Persistent Therapy During 12 Months Post-index Date
Description: Index medication persistent therapy duration was defined as days to discontinue or immediate switch or end of 12 months post-index follow if participants remained persistent, whichever came first. Index medications were tofacitinib, adalimumab or etanercept. Persistent with the index medication: not having a gap in the therapy of at least 60 days between prescription fill dates and their administration. Discontinuation from index medication: gap in the index medication therapy of at least 60 days. Immediate switch from index medication: initiation of a non-index advanced therapy before end of a 60-day gap in index medication.
Time Frame: During 12 months post-index date
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Tofacitinib Low OOP Cost | Tofacitinib High OOP Cost | Switch From Adalimumab to Etanercept | Switch From Adalimumab to Tofacitinib | Switch From Etanercept to Adalimumab | Switch From Etanercept to Tofacitinib
Number analyzed (Participants) | 310 | 299 | 79 | 287 | 112 | 262
Days | 235.60 (133.02) | 273.50 (136.81) | 203.65 (133.21) | 239.02 (134.51) | 219.75 (126.09) | 234.34 (131.10)
Statistical Analysis 1: Comparison: Tofacitinib Low OOP Cost vs Tofacitinib High OOP Cost; Test type: Superiority; p = 0.1736, Log Rank
Statistical Analysis 2: Comparison: Switch From Adalimumab to Etanercept vs Switch From Adalimumab to Tofacitinib; Test type: Superiority; p = 0.0195, Log Rank
Statistical Analysis 3: Comparison: Switch From Etanercept to Adalimumab vs Switch From Etanercept to Tofacitinib; Test type: Superiority; p = 0.2104, Log Rank
Statistical Analysis 4: Comparison: Tofacitinib Low OOP Cost vs Tofacitinib High OOP Cost; [analysis description as in outcome 1, analysis 4]; Test type: Superiority; p = 0.1670, Regression, Cox; Hazard Ratio (HR) = 1.1723, 95% CI 2-sided [0.9357 to 1.4687]
Statistical Analysis 5: Comparison: Switch From Adalimumab to Etanercept vs Switch From Adalimumab to Tofacitinib; [analysis description as in outcome 1, analysis 4]; Test type: Superiority; p = 0.1087, Regression, Cox; Hazard Ratio (HR) = 0.7228, 95% CI 2-sided [0.4861 to 1.0747]
Statistical Analysis 6: Comparison: Switch From Etanercept to Adalimumab vs Switch From Etanercept to Tofacitinib; [analysis description as in outcome 1, analysis 4]; Test type: Superiority; p = 0.3212, Regression, Cox; Hazard Ratio (HR) = 0.8402, 95% CI 2-sided [0.5957 to 1.1852]

11. Secondary Outcome: Percentage of Participants Who Were Persistent With Main Non-Biologic Disease Modifying Antirheumatic Drugs (NB-DMARD) During 12 Months Post-index Date: Combination Therapy
Description: Participants who initiated index medication in combination with main NB-DMARDSs were analyzed to evaluate percentage of participants who were persistent with main NB-DMARDs use. Main NB-DMARDs considered in the study were methotrexate, sulfasalazine, leflunomide, and hydroxychloroquine. Index medications were tofacitinib, adalimumab or etanercept. Persistence with main NB-DMARDs was defined as not having a gap of at least 60 days between prescription fill dates and their administration.
Time Frame: During 12 months post-index date
Population: as for outcome 7
Measure: Number; unit: Percentage of participants
Arm/Group | Tofacitinib Low OOP Cost | Tofacitinib High OOP Cost | Switch From Adalimumab to Etanercept | Switch From Adalimumab to Tofacitinib | Switch From Etanercept to Adalimumab | Switch From Etanercept to Tofacitinib
Number analyzed (Participants) | 157 | 145 | 44 | 151 | 57 | 105
Percentage of participants | 36.31 | 35.86 | 36.36 | 43.71 | 38.60 | 42.86
Statistical Analysis 1: Comparison: Tofacitinib Low OOP Cost vs Tofacitinib High OOP Cost; Test type: Superiority; p = 0.9361, Chi-squared
Statistical Analysis 2: Comparison: Switch From Adalimumab to Etanercept vs Switch From Adalimumab to Tofacitinib; Test type: Superiority; p = 0.3851, Chi-squared
Statistical Analysis 3: Comparison: Switch From Etanercept to Adalimumab vs Switch From Etanercept to Tofacitinib; Test type: Superiority; p = 0.5990, Chi-squared
Statistical Analysis 4: Comparison: Tofacitinib Low OOP Cost vs Tofacitinib High OOP Cost; [analysis description as in outcome 1, analysis 4]; Test type: Superiority; p = 0.9860, Regression, Logistic; Odds Ratio (OR) = 0.9954, 95% CI 2-sided [0.5962 to 1.6620]
Statistical Analysis 5: Comparison: Switch From Adalimumab to Etanercept vs Switch From Adalimumab to Tofacitinib; [analysis description as in outcome 1, analysis 4]; Test type: Superiority; p = 0.5813, Regression, Logistic; Odds Ratio (OR) = 1.2959, 95% CI 2-sided [0.5158 to 3.2558]
Statistical Analysis 6: Comparison: Switch From Etanercept to Adalimumab vs Switch From Etanercept to Tofacitinib; To control and remove the possible influence of the independent variables (like treatment cohort, demographic and clinical characteristics of interest, etc. and clinical judgement) on the outcome measure, multivariable analysis was performed; Test type: Superiority; p = 0.1789, Regression, Logistic; Odds Ratio (OR) = 1.8182, 95% CI 2-sided [0.7604 to 4.3473]

12. Secondary Outcome: Percentage of Participants Who Immediately Switched From Main NB-DMARDs During 12 Months Post-index Date: Combination Therapy
Description: Participants who initiated index medication in combination with main NB-DMARDSs were analyzed to evaluate percentage of participants who immediately switched from main NB-DMARDs. Main NB-DMARDS considered in the study were methotrexate, sulfasalazine, leflunomide, and hydroxychloroquine. Index medications were tofacitinib, adalimumab or etanercept. Immediate switch from main NB-DMARDs was defined as initiation of other medication than main NB-DMARDs, before end of a 60-day gap.
Time Frame: During 12 months post-index date
Population: as for outcome 7
Measure: Number; unit: Percentage of participants
Arm/Group | Tofacitinib Low OOP Cost | Tofacitinib High OOP Cost | Switch From Adalimumab to Etanercept | Switch From Adalimumab to Tofacitinib | Switch From Etanercept to Adalimumab | Switch From Etanercept to Tofacitinib
Number analyzed (Participants) | 157 | 145 | 44 | 151 | 57 | 105
Percentage of participants | 30.57 | 26.21 | 22.73 | 22.52 | 31.58 | 23.81
Statistical Analysis 1: Comparison: Tofacitinib Low OOP Cost vs Tofacitinib High OOP Cost; Test type: Superiority; p = 0.4009, Chi-squared
Statistical Analysis 2: Comparison: Switch From Adalimumab to Etanercept vs Switch From Adalimumab to Tofacitinib; Test type: Superiority; p = 0.9765, Chi-squared
Statistical Analysis 3: Comparison: Switch From Etanercept to Adalimumab vs Switch From Etanercept to Tofacitinib; Test type: Superiority; p = 0.2849, Chi-squared
Statistical Analysis 4: Comparison: Tofacitinib Low OOP Cost vs Tofacitinib High OOP Cost; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p = 0.5289, Regression, Logistic; Odds Ratio (OR) = 0.8252, 95% CI 2-sided [0.4538 to 1.5007]
Statistical Analysis 5: Comparison: Switch From Adalimumab to Etanercept vs Switch From Adalimumab to Tofacitinib; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p = 0.9270, Regression, Logistic; Odds Ratio (OR) = 0.9408, 95% CI 2-sided [0.2553 to 3.4678]
Statistical Analysis 6: Comparison: Switch From Etanercept to Adalimumab vs Switch From Etanercept to Tofacitinib; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p = 0.0707, Regression, Logistic; Odds Ratio (OR) = 0.3968, 95% CI 2-sided [0.1456 to 1.0812]

13. Secondary Outcome: Percentage of Participants Who Discontinued Then Switched From Main NB-DMARDs During 12 Months Post-index Date: Combination Therapy
Description: Participants who initiated index medication in combination with main NB-DMARDSs were analyzed to evaluate percentage of participants who discontinued then switched from main NB-DMARDs. Main NB-DMARDS considered in the study were methotrexate, sulfasalazine, leflunomide, and hydroxychloroquine. Index medications were tofacitinib, adalimumab or etanercept. Participants who discontinued main NB-DMARDs then switched from main NB-DMARDS were those who had gap in the main NB-DMARDs medication of at least 60 days and then after the gap switched to other medication than main NB-DMARDs.
Time Frame: During 12 months post-index date
Population: as for outcome 7
Measure: Number; unit: Percentage of participants
Arm/Group | Tofacitinib Low OOP Cost | Tofacitinib High OOP Cost | Switch From Adalimumab to Etanercept | Switch From Adalimumab to Tofacitinib | Switch From Etanercept to Adalimumab | Switch From Etanercept to Tofacitinib
Number analyzed (Participants) | 157 | 145 | 44 | 151 | 57 | 105
Percentage of participants | 2.55 | 0.69 | 6.82 | 2.65 | 0.00 | 0.00
Statistical Analysis 1: Comparison: Tofacitinib Low OOP Cost vs Tofacitinib High OOP Cost; Test type: Superiority; p = 0.2061, Chi-squared
Statistical Analysis 2: Comparison: Switch From Adalimumab to Etanercept vs Switch From Adalimumab to Tofacitinib; Test type: Superiority; p = 0.1908, Chi-squared

14. Secondary Outcome: Percentage of Participants Who Discontinued Then Restarted Main NB-DMARDs During 12 Months Post-index Date: Combination Therapy
Description: Participants who initiated index medication in combination with main NB-DMARDSs were analyzed to evaluate percentage of participants who discontinued then restarted main NB-DMARDs. Main NB-DMARDS considered in the study were methotrexate, sulfasalazine, leflunomide, and hydroxychloroquine. Index medications were tofacitinib, adalimumab or etanercept. Participants who discontinued main NB-DMARDs and then restarted main NB-DMARDs were those who had a gap in main NB-DMARDs of at least 60 days and after the gap, they started main NB-DMARDs again.
Time Frame: During 12 months post-index date
Population: as for outcome 7
Measure: Number; unit: Percentage of participants
Arm/Group | Tofacitinib Low OOP Cost | Tofacitinib High OOP Cost | Switch From Adalimumab to Etanercept | Switch From Adalimumab to Tofacitinib | Switch From Etanercept to Adalimumab | Switch From Etanercept to Tofacitinib
Number analyzed (Participants) | 157 | 145 | 44 | 151 | 57 | 105
Percentage of participants | 13.38 | 12.41 | 13.64 | 11.26 | 21.05 | 18.10
Statistical Analysis 1: Comparison: Tofacitinib Low OOP Cost vs Tofacitinib High OOP Cost; Test type: Superiority; p = 0.8033, Chi-squared
Statistical Analysis 2: Comparison: Switch From Adalimumab to Etanercept vs Switch From Adalimumab to Tofacitinib; Test type: Superiority; p = 0.6669, Chi-squared
Statistical Analysis 3: Comparison: Switch From Etanercept to Adalimumab vs Switch From Etanercept to Tofacitinib; Test type: Superiority; p = 0.6477, Chi-squared
Statistical Analysis 4: Comparison: Tofacitinib Low OOP Cost vs Tofacitinib High OOP Cost; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p = 0.5509, Regression, Logistic; Odds Ratio (OR) = 0.7948, 95% CI 2-sided [0.3736 to 1.6907]
Statistical Analysis 5: Comparison: Switch From Adalimumab to Etanercept vs Switch From Adalimumab to Tofacitinib; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p = 0.6216, Regression, Logistic; Odds Ratio (OR) = 0.6814, 95% CI 2-sided [0.1486 to 3.1250]
Statistical Analysis 6: Comparison: Switch From Etanercept to Adalimumab vs Switch From Etanercept to Tofacitinib; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p = 0.5506, Regression, Logistic; Odds Ratio (OR) = 0.6974, 95% CI 2-sided [0.2135 to 2.2781]

15. Secondary Outcome: Percentage of Participants Who Discontinued Without Switching or Restarting Main NB-DMARDs During 12 Months Post-index Date: Combination Therapy
Description: Participants who initiated index medication in combination with main NB-DMARDSs were analyzed to evaluate percentage of participants who discontinued without switching or restarting main NB-DMARDs. Main NB-DMARDS considered in the study were methotrexate, sulfasalazine, leflunomide, and hydroxychloroquine. Index medications were tofacitinib, adalimumab or etanercept. Participants who discontinued main NB-DMARDs without switching or restarting main NB-DMARDs were those who had a gap in main NB-DMARDs of at least 60 days and there were no claims for either the main NB-DMARDs or a different therapy for the remainder of the follow-up period.
Time Frame: During 12 months post-index date
Population: as for outcome 7
Measure: Number; unit: Percentage of participants
Arm/Group | Tofacitinib Low OOP Cost | Tofacitinib High OOP Cost | Switch From Adalimumab to Etanercept | Switch From Adalimumab to Tofacitinib | Switch From Etanercept to Adalimumab | Switch From Etanercept to Tofacitinib
Number analyzed (Participants) | 157 | 145 | 44 | 151 | 57 | 105
Percentage of participants | 17.20 | 24.83 | 20.45 | 19.87 | 8.77 | 15.24
Statistical Analysis 1: Comparison: Tofacitinib Low OOP Cost vs Tofacitinib High OOP Cost; Test type: Superiority; p = 0.1030, Chi-squared
Statistical Analysis 2: Comparison: Switch From Adalimumab to Etanercept vs Switch From Adalimumab to Tofacitinib; Test type: Superiority; p = 0.9317, Chi-squared
Statistical Analysis 3: Comparison: Switch From Etanercept to Adalimumab vs Switch From Etanercept to Tofacitinib; Test type: Superiority; p = 0.2420, Chi-squared
Statistical Analysis 4: Comparison: Tofacitinib Low OOP Cost vs Tofacitinib High OOP Cost; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p = 0.0869, Regression, Logistic; Odds Ratio (OR) = 1.7474, 95% CI 2-sided [0.9222 to 3.3107]
Statistical Analysis 5: Comparison: Switch From Adalimumab to Etanercept vs Switch From Adalimumab to Tofacitinib; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p = 0.8228, Regression, Logistic; Odds Ratio (OR) = 1.1346, 95% CI 2-sided [0.3757 to 3.4266]
Statistical Analysis 6: Comparison: Switch From Etanercept to Adalimumab vs Switch From Etanercept to Tofacitinib; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p = 0.4855, Regression, Logistic; Odds Ratio (OR) = 1.5650, 95% CI 2-sided [0.4446 to 5.5086]

16. Secondary Outcome: Percentage of Participants Who Initiated Index Medication as Monotherapy and Eventually Added NB-DMARDs During 12 Months Post-index Date
Description: Percentage of participants who initiated only index medication and then eventually also added any NB-DMARDs, 1 of the 4 mains NB-DMARDs or other than these 4 NB-DMARDs in their therapy, were evaluated. Main NB-DMARDS considered in the study were methotrexate, sulfasalazine, leflunomide, and hydroxychloroquine. Any NB-DMARDs included those participants who received any of the NB-DMARDs and participant was counted only once if took different NB-DMARDs during the follow-up period. Participants might be counted more than once in categories except category "Any NB-DMARDs". Index medications were tofacitinib, adalimumab or etanercept.
Time Frame: During 12 months post-index date
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | Tofacitinib Low OOP Cost | Tofacitinib High OOP Cost | Switch From Adalimumab to Etanercept | Switch From Adalimumab to Tofacitinib | Switch From Etanercept to Adalimumab | Switch From Etanercept to Tofacitinib
Number analyzed (Participants) | 310 | 299 | 79 | 287 | 112 | 262
Percentage of participants
  Any NB-DMARD | 29.41 | 28.57 | 48.57 | 25.74 | 34.55 | 26.75
  Methotrexate | 16.99 | 11.69 | 22.86 | 14.71 | 27.27 | 12.74
  Sulfasalazine | 1.96 | 2.60 | 8.57 | 2.21 | 5.45 | 1.91
  Leflunomide | 3.92 | 5.19 | 17.14 | 5.15 | 3.64 | 6.37
  Hydroxychloroquine | 8.50 | 9.09 | 20.00 | 3.68 | 5.45 | 5.10
  Other NB-DMARD | 3.27 | 3.90 | 2.86 | 1.47 | 0.00 | 4.46

17. Secondary Outcome: Percentage of Participants Who Met Adherence Effectiveness Criteria During 12 Months Post-index Date
Description: A proportion of days covered (PDC) was calculated based on total days' supply over the 12 months post-index. The PDC was calculated by using the date of service and the day supply for each fill of the index medication. Participants with early refills were allowed to stockpile medications up to a maximum of 14 days total for later use. Participants who met adherence effective criteria were those who had PDC >=0.8. Index medications were tofacitinib, adalimumab or etanercept.
Time Frame: During 12 months post-index date
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | Tofacitinib Low OOP Cost | Tofacitinib High OOP Cost | Switch From Adalimumab to Etanercept | Switch From Adalimumab to Tofacitinib | Switch From Etanercept to Adalimumab | Switch From Etanercept to Tofacitinib
Number analyzed (Participants) | 310 | 299 | 79 | 287 | 112 | 262
Percentage of participants | 38.71 | 36.12 | 30.38 | 44.95 | 33.04 | 38.93
Statistical Analysis 1: Comparison: Tofacitinib Low OOP Cost vs Tofacitinib High OOP Cost; Test type: Superiority; p = 0.5092, Chi-squared
Statistical Analysis 2: Comparison: Switch From Adalimumab to Etanercept vs Switch From Adalimumab to Tofacitinib; Test type: Superiority; p = 0.0201, Chi-squared
Statistical Analysis 3: Comparison: Switch From Etanercept to Adalimumab vs Switch From Etanercept to Tofacitinib; Test type: Superiority; p = 0.2799, Chi-squared
Statistical Analysis 4: Comparison: Tofacitinib Low OOP Cost vs Tofacitinib High OOP Cost; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p = 0.5772, Regression, Logistic; Odds Ratio (OR) = 0.9021, 95% CI 2-sided [0.6281 to 1.2958]
Statistical Analysis 5: Comparison: Switch From Adalimumab to Etanercept vs Switch From Adalimumab to Tofacitinib; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p = 0.3272, Regression, Logistic; Odds Ratio (OR) = 1.3953, 95% CI 2-sided [0.7166 to 2.7169]
Statistical Analysis 6: Comparison: Switch From Etanercept to Adalimumab vs Switch From Etanercept to Tofacitinib; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p = 0.3011, Regression, Logistic; Odds Ratio (OR) = 1.3527, 95% CI 2-sided [0.7630 to 2.3983]

18. Secondary Outcome: Percentage of Participants Who Met Dose Escalation Effectiveness Criteria During 12 Months Post-index Date
Description: Dose escalation for index medication was defined as: 1) for adalimumab: at least 1 claim in the 12 months post-index follow-up with an average weekly dose of at least 40 milligram per week (mg/week), 2) for etanercept: at least 1 claim in the 12 months post-index follow-up with an average weekly dose of at least 100 mg/week, 3) for tofacitinib: at least 1 claim in the 12 months post-index follow-up with an average weekly dose of at least 20 milligram per day (mg/day) for immediate release and 22 mg/day for extended release. Participants who met dose escalation effectiveness criteria were those who did not have any dose escalation for index medication compared to the starting dose.
Time Frame: During 12 months post-index date
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | Tofacitinib Low OOP Cost | Tofacitinib High OOP Cost | Switch From Adalimumab to Etanercept | Switch From Adalimumab to Tofacitinib | Switch From Etanercept to Adalimumab | Switch From Etanercept to Tofacitinib
Number analyzed (Participants) | 310 | 299 | 79 | 287 | 112 | 262
Percentage of participants | 96.13 | 94.31 | 97.47 | 94.77 | 81.25 | 95.80
Statistical Analysis 1: Comparison: Tofacitinib Low OOP Cost vs Tofacitinib High OOP Cost; Test type: Superiority; p = 0.2931, Chi-squared
Statistical Analysis 2: Comparison: Switch From Adalimumab to Etanercept vs Switch From Adalimumab to Tofacitinib; Test type: Superiority; p = 0.3135, Chi-squared
Statistical Analysis 3: Comparison: Switch From Etanercept to Adalimumab vs Switch From Etanercept to Tofacitinib; Test type: Superiority; p < 0.0001, Chi-squared
Statistical Analysis 4: Comparison: Tofacitinib Low OOP Cost vs Tofacitinib High OOP Cost; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p = 0.6772, Regression, Logistic; Odds Ratio (OR) = 0.8369, 95% CI 2-sided [0.3618 to 1.9356]
Statistical Analysis 5: Comparison: Switch From Etanercept to Adalimumab vs Switch From Etanercept to Tofacitinib; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p = 0.0013, Regression, Logistic; Odds Ratio (OR) = 5.2530, 95% CI 2-sided [1.9061 to 14.4770]

19. Secondary Outcome: Percentage of Participants Who Met Switched Effectiveness Criteria During 12 Months Post-index Date
Description: A switch for this outcome measure was defined as use of a different biologic disease modifying antirheumatic drug (B-DMARDs) or Janus kinase inhibitor (JAKi), any time during the 12 months post-index follow-up. Participants who met switched effectiveness criteria were those who did not switch from the index medication to B-DMARDs or JAKi. Index medications were tofacitinib, adalimumab or etanercept.
Time Frame: During 12 months post-index date
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | Tofacitinib Low OOP Cost | Tofacitinib High OOP Cost | Switch From Adalimumab to Etanercept | Switch From Adalimumab to Tofacitinib | Switch From Etanercept to Adalimumab | Switch From Etanercept to Tofacitinib
Number analyzed (Participants) | 310 | 299 | 79 | 287 | 112 | 262
Percentage of participants | 85.81 | 83.95 | 65.82 | 77.00 | 64.29 | 70.23
Statistical Analysis 1: Comparison: Tofacitinib Low OOP Cost vs Tofacitinib High OOP Cost; Test type: Superiority; p = 0.5217, Chi-squared
Statistical Analysis 2: Comparison: Switch From Adalimumab to Etanercept vs Switch From Adalimumab to Tofacitinib; Test type: Superiority; p = 0.0432, Chi-squared
Statistical Analysis 3: Comparison: Switch From Etanercept to Adalimumab vs Switch From Etanercept to Tofacitinib; Test type: Superiority; p = 0.2573, Chi-squared
Statistical Analysis 4: Comparison: Tofacitinib Low OOP Cost vs Tofacitinib High OOP Cost; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p = 0.5368, Regression, Logistic; Odds Ratio (OR) = 0.8593, 95% CI 2-sided [0.5311 to 1.3902]
Statistical Analysis 5: Comparison: Switch From Adalimumab to Etanercept vs Switch From Adalimumab to Tofacitinib; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p = 0.4685, Regression, Logistic; Odds Ratio (OR) = 1.2892, 95% CI 2-sided [0.6488 to 2.5616]
Statistical Analysis 6: Comparison: Switch From Etanercept to Adalimumab vs Switch From Etanercept to Tofacitinib; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p = 0.3112, Regression, Logistic; Odds Ratio (OR) = 1.3598, 95% CI 2-sided [0.7502 to 2.4648]

20. Secondary Outcome: Percentage of Participants Who Met NB-DMARD Effectiveness Criteria During 12 Months Post-index Date
Description: Participants who started only index medication regimen (as monotherapy), but eventually initiated main NB-DMARDs were identified in the 12 months post-index follow-up period as adding new NB-DMARD. Participants who started index medication regimen along with any of the main NB-DMARDs (combination therapy), presence of a different NB-DMARD in 12 months post-index was identified as adding new NB-DMARD. Participants who met NB-DMARD effectiveness criteria were those who did not add a new NB-DMARD in the 12 months post-index follow up. Index medications were tofacitinib, adalimumab or etanercept.
Time Frame: During 12 months post-index date
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | Tofacitinib Low OOP Cost | Tofacitinib High OOP Cost | Switch From Adalimumab to Etanercept | Switch From Adalimumab to Tofacitinib | Switch From Etanercept to Adalimumab | Switch From Etanercept to Tofacitinib
Number analyzed (Participants) | 310 | 299 | 79 | 287 | 112 | 262
Percentage of participants | 71.61 | 74.58 | 64.56 | 77.00 | 66.96 | 79.39
Statistical Analysis 1: Comparison: Tofacitinib Low OOP Cost vs Tofacitinib High OOP Cost; Test type: Superiority; p = 0.4090, Chi-squared
Statistical Analysis 2: Comparison: Switch From Adalimumab to Etanercept vs Switch From Adalimumab to Tofacitinib; Test type: Superiority; p = 0.0249, Chi-squared
Statistical Analysis 3: Comparison: Switch From Etanercept to Adalimumab vs Switch From Etanercept to Tofacitinib; Test type: Superiority; p = 0.0103, Chi-squared
Statistical Analysis 4: Comparison: Tofacitinib Low OOP Cost vs Tofacitinib High OOP Cost; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p = 0.5415, Regression, Logistic; Odds Ratio (OR) = 1.1302, 95% CI 2-sided [0.7630 to 1.6741]
Statistical Analysis 5: Comparison: Switch From Adalimumab to Etanercept vs Switch From Adalimumab to Tofacitinib; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p = 0.0596, Regression, Logistic; Odds Ratio (OR) = 2.0118, 95% CI 2-sided [0.9722 to 4.1632]
Statistical Analysis 6: Comparison: Switch From Etanercept to Adalimumab vs Switch From Etanercept to Tofacitinib; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p = 0.0002, Regression, Logistic; Odds Ratio (OR) = 3.4823, 95% CI 2-sided [1.7930 to 6.7633]

21. Secondary Outcome: Percentage of Participants Who Met Oral Glucocorticoid Effectiveness Criteria During 12 Months Post-index Date
Description: Oral glucocorticoid effectiveness criteria for participants with no claims for oral glucocorticoid prescriptions in the 6 months prior to the index date = did not receive more than 30 days of oral glucocorticoids between (index date + 89 days) to (index date + 359 days). 30 days of oral glucocorticoids was determined by summing up the day supply of all glucocorticoids claims with a fill date between (index date + 89 days) to (index date + 359 days). Oral glucocorticoid effectiveness criteria for participants with claims for oral glucocorticoids during the 6 months prior to the index date = no increase in oral glucocorticoid dose >=20% during months 6-12 after index compared to the 6 months before the index date. Increase in oral glucocorticoids was determined from the prednisone equivalent dose for all glucocorticoid claims filled.
Time Frame: During 12 months post-index date
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | Tofacitinib Low OOP Cost | Tofacitinib High OOP Cost | Switch From Adalimumab to Etanercept | Switch From Adalimumab to Tofacitinib | Switch From Etanercept to Adalimumab | Switch From Etanercept to Tofacitinib
Number analyzed (Participants) | 310 | 299 | 79 | 287 | 112 | 262
Percentage of participants | 83.55 | 86.96 | 83.54 | 85.02 | 86.61 | 81.30
Statistical Analysis 1: Comparison: Tofacitinib Low OOP Cost vs Tofacitinib High OOP Cost; Test type: Superiority; p = 0.2361, Chi-squared
Statistical Analysis 2: Comparison: Switch From Adalimumab to Etanercept vs Switch From Adalimumab to Tofacitinib; Test type: Superiority; p = 0.7474, Chi-squared
Statistical Analysis 3: Comparison: Switch From Etanercept to Adalimumab vs Switch From Etanercept to Tofacitinib; Test type: Superiority; p = 0.2118, Chi-squared
Statistical Analysis 4: Comparison: Tofacitinib Low OOP Cost vs Tofacitinib High OOP Cost; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p = 0.1978, Regression, Logistic; Odds Ratio (OR) = 1.3811, 95% CI 2-sided [0.8449 to 2.2576]
Statistical Analysis 5: Comparison: Switch From Adalimumab to Etanercept vs Switch From Adalimumab to Tofacitinib; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p = 0.8893, Regression, Logistic; Odds Ratio (OR) = 1.0614, 95% CI 2-sided [0.4587 to 2.4559]
Statistical Analysis 6: Comparison: Switch From Etanercept to Adalimumab vs Switch From Etanercept to Tofacitinib; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p = 0.1553, Regression, Logistic; Odds Ratio (OR) = 0.5811, 95% CI 2-sided [0.2748 to 1.2286]

22. Secondary Outcome: Percentage of Participants Who Met Infusion Glucocorticoid Effectiveness Criteria During 12 Months Post-index Date
Description: Glucocorticoid infusion effectiveness criteria was receiving of maximum of 1 parenteral or intra-articular glucocorticoid joint injection on unique days (between [index date + 89 days] to [index date + 359 days]) after the participants had been on treatment with index medication for more than 3 months. Index medications were tofacitinib, adalimumab or etanercept.
Time Frame: During 12 months post-index date
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | Tofacitinib Low OOP Cost | Tofacitinib High OOP Cost | Switch From Adalimumab to Etanercept | Switch From Adalimumab to Tofacitinib | Switch From Etanercept to Adalimumab | Switch From Etanercept to Tofacitinib
Number analyzed (Participants) | 310 | 299 | 79 | 287 | 112 | 262
Percentage of participants | 83.87 | 82.61 | 74.68 | 82.58 | 83.04 | 76.34
Statistical Analysis 1: Comparison: Tofacitinib Low OOP Cost vs Tofacitinib High OOP Cost; Test type: Superiority; p = 0.6767, Chi-squared
Statistical Analysis 2: Comparison: Switch From Adalimumab to Etanercept vs Switch From Adalimumab to Tofacitinib; Test type: Superiority; p = 0.1141, Chi-squared
Statistical Analysis 3: Comparison: Switch From Etanercept to Adalimumab vs Switch From Etanercept to Tofacitinib; Test type: Superiority; p = 0.1497, Chi-squared
Statistical Analysis 4: Comparison: Tofacitinib Low OOP Cost vs Tofacitinib High OOP Cost; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p = 0.5228, Regression, Logistic; Odds Ratio (OR) = 0.8556, 95% CI 2-sided [0.5303 to 1.3804]
Statistical Analysis 5: Comparison: Switch From Adalimumab to Etanercept vs Switch From Adalimumab to Tofacitinib; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p = 0.0277, Regression, Logistic; Odds Ratio (OR) = 2.5125, 95% CI 2-sided [1.1062 to 5.7063]
Statistical Analysis 6: Comparison: Switch From Etanercept to Adalimumab vs Switch From Etanercept to Tofacitinib; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p = 0.3240, Regression, Logistic; Odds Ratio (OR) = 0.6993, 95% CI 2-sided [0.3435 to 1.4236]

23. Secondary Outcome: Mean of Rheumatoid Arthritis (RA) Related Inpatient Visits During 12 Months Pre-index Date
Description: Inpatient visits refers when participants visited hospital for formal admission. In this outcome measure, mean of number of inpatient visits related to RA during 12 months pre-index were evaluated.
Time Frame: During 12 months pre-index date
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Inpatient visits
Arm/Group | Tofacitinib Low OOP Cost | Tofacitinib High OOP Cost | Switch From Adalimumab to Etanercept | Switch From Adalimumab to Tofacitinib | Switch From Etanercept to Adalimumab | Switch From Etanercept to Tofacitinib
Number analyzed (Participants) | 310 | 299 | 79 | 287 | 112 | 262
Inpatient visits | 0.08 (0.28) | 0.09 (0.38) | 0.05 (0.22) | 0.08 (0.31) | 0.04 (0.25) | 0.08 (0.32)
Statistical Analysis 1: Comparison: Tofacitinib Low OOP Cost vs Tofacitinib High OOP Cost; Test type: Superiority; p = 0.6318, t-test, 2 sided
Statistical Analysis 2: Comparison: Switch From Adalimumab to Etanercept vs Switch From Adalimumab to Tofacitinib; Test type: Superiority; p = 0.3802, t-test, 2 sided
Statistical Analysis 3: Comparison: Switch From Etanercept to Adalimumab vs Switch From Etanercept to Tofacitinib; Test type: Superiority; p = 0.2424, t-test, 2 sided
Statistical Analysis 4: Comparison: Tofacitinib Low OOP Cost vs Tofacitinib High OOP Cost; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p = 0.1753, Regression, Linear; Odds Ratio (OR) = 0.0347, 95% CI 2-sided [-0.0155 to 0.0848]
Statistical Analysis 5: Comparison: Switch From Adalimumab to Etanercept vs Switch From Adalimumab to Tofacitinib; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p = 0.6114, Regression, Linear; Odds Ratio (OR) = 0.0194, 95% CI 2-sided [-0.0553 to 0.0941]
Statistical Analysis 6: Comparison: Switch From Etanercept to Adalimumab vs Switch From Etanercept to Tofacitinib; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p = 0.2977, Regression, Linear; Odds Ratio (OR) = 0.0345, 95% CI 2-sided [-0.0304 to 0.0993]

24. Secondary Outcome: Mean of Rheumatoid Arthritis Related Emergency Department (ED) Visits During 12 Months Pre-Index Date
Description: In this outcome measure, mean of number of emergency department visits related to RA during 12 months pre-index were evaluated.
Time Frame: During 12 months pre-index date
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Emergency department visits
Arm/Group | Tofacitinib Low OOP Cost | Tofacitinib High OOP Cost | Switch From Adalimumab to Etanercept | Switch From Adalimumab to Tofacitinib | Switch From Etanercept to Adalimumab | Switch From Etanercept to Tofacitinib
Number analyzed (Participants) | 310 | 299 | 79 | 287 | 112 | 262
Emergency department visits | 0.16 (0.53) | 0.10 (0.44) | 0.13 (0.54) | 0.14 (0.44) | 0.14 (0.75) | 0.21 (0.94)
Statistical Analysis 1: Comparison: Tofacitinib Low OOP Cost vs Tofacitinib High OOP Cost; Test type: Superiority; p = 0.1473, t-test, 2 sided
Statistical Analysis 2: Comparison: Switch From Adalimumab to Etanercept vs Switch From Adalimumab to Tofacitinib; Test type: Superiority; p = 0.8747, t-test, 2 sided
Statistical Analysis 3: Comparison: Switch From Etanercept to Adalimumab vs Switch From Etanercept to Tofacitinib; Test type: Superiority; p = 0.5265, t-test, 2 sided
Statistical Analysis 4: Comparison: Tofacitinib Low OOP Cost vs Tofacitinib High OOP Cost; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p = 0.2522, Regression, Linear; Odds Ratio (OR) = -0.0457, 95% CI 2-sided [-0.1239 to 0.0325]
Statistical Analysis 5: Comparison: Switch From Adalimumab to Etanercept vs Switch From Adalimumab to Tofacitinib; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p = 0.6701, Regression, Linear; Odds Ratio (OR) = 0.0278, 95% CI 2-sided [-0.1003 to 0.1559]
Statistical Analysis 6: Comparison: Switch From Etanercept to Adalimumab vs Switch From Etanercept to Tofacitinib; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p = 0.1017, Regression, Linear; Odds Ratio (OR) = 0.1693, 95% CI 2-sided [-0.0334 to 0.3720]

25. Secondary Outcome: Mean of Rheumatoid Arthritis Related Outpatient Visits During 12 Months Pre-index Date
Description: Outpatient visits refers when participants visited hospital but not for formal admission. In this outcome measure, mean of number of outpatient visits related to RA during 12 months pre-index were evaluated.
Time Frame: During 12 months pre-index date
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Outpatient visits
Arm/Group | Tofacitinib Low OOP Cost | Tofacitinib High OOP Cost | Switch From Adalimumab to Etanercept | Switch From Adalimumab to Tofacitinib | Switch From Etanercept to Adalimumab | Switch From Etanercept to Tofacitinib
Number analyzed (Participants) | 310 | 299 | 79 | 287 | 112 | 262
Outpatient visits | 7.83 (5.69) | 8.38 (5.45) | 7.90 (5.54) | 8.80 (5.66) | 7.19 (4.61) | 8.89 (5.22)
Statistical Analysis 1: Comparison: Tofacitinib Low OOP Cost vs Tofacitinib High OOP Cost; Test type: Superiority; p = 0.2246, t-test, 2 sided
Statistical Analysis 2: Comparison: Switch From Adalimumab to Etanercept vs Switch From Adalimumab to Tofacitinib; Test type: Superiority; p = 0.2101, t-test, 2 sided
Statistical Analysis 3: Comparison: Switch From Etanercept to Adalimumab vs Switch From Etanercept to Tofacitinib; Test type: Superiority; p = 0.0030, t-test, 2 sided
Statistical Analysis 4: Comparison: Tofacitinib Low OOP Cost vs Tofacitinib High OOP Cost; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p = 0.3324, Regression, Linear; Odds Ratio (OR) = 0.4140, 95% CI 2-sided [-0.4231 to 1.2511]
Statistical Analysis 5: Comparison: Switch From Adalimumab to Etanercept vs Switch From Adalimumab to Tofacitinib; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p = 0.1367, Regression, Linear; Odds Ratio (OR) = 1.1712, 95% CI 2-sided [-0.3713 to 2.7138]
Statistical Analysis 6: Comparison: Switch From Etanercept to Adalimumab vs Switch From Etanercept to Tofacitinib; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p = 0.0028, Regression, Linear; Odds Ratio (OR) = 1.8099, 95% CI 2-sided [0.6219 to 2.9978]

26. Secondary Outcome: Mean of Rheumatoid Arthritis-Related Pharmacy Visits During 12 Months Pre-index Date
Description: In this outcome measure, mean of number of pharmacy visits related to RA during 12 months pre-index were evaluated.
Time Frame: During 12 months pre-index date
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Pharmacy visits
Arm/Group | Tofacitinib Low OOP Cost | Tofacitinib High OOP Cost | Switch From Adalimumab to Etanercept | Switch From Adalimumab to Tofacitinib | Switch From Etanercept to Adalimumab | Switch From Etanercept to Tofacitinib
Number analyzed (Participants) | 310 | 299 | 79 | 287 | 112 | 262
Pharmacy visits | 13.25 (9.80) | 14.16 (10.45) | 17.23 (11.53) | 17.85 (10.80) | 16.60 (11.18) | 17.40 (11.69)
Statistical Analysis 1: Comparison: Tofacitinib Low OOP Cost vs Tofacitinib High OOP Cost; Test type: Superiority; p = 0.2667, t-test, 2 sided
Statistical Analysis 2: Comparison: Switch From Adalimumab to Etanercept vs Switch From Adalimumab to Tofacitinib; Test type: Superiority; p = 0.6570, t-test, 2 sided
Statistical Analysis 3: Comparison: Switch From Etanercept to Adalimumab vs Switch From Etanercept to Tofacitinib; Test type: Superiority; p = 0.5403, t-test, 2 sided
Statistical Analysis 4: Comparison: Tofacitinib Low OOP Cost vs Tofacitinib High OOP Cost; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p = 0.1167, Regression, Linear; Odds Ratio (OR) = 0.9159, 95% CI 2-sided [-0.2283 to 2.0600]
Statistical Analysis 5: Comparison: Switch From Adalimumab to Etanercept vs Switch From Adalimumab to Tofacitinib; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p = 0.9722, Regression, Linear; Odds Ratio (OR) = -0.0336, 95% CI 2-sided [-1.9238 to 1.8567]
Statistical Analysis 6: Comparison: Switch From Etanercept to Adalimumab vs Switch From Etanercept to Tofacitinib; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p = 0.8455, Regression, Logistic; Odds Ratio (OR) = 0.2064, 95% CI 2-sided [-1.8689 to 2.2817]

27. Secondary Outcome: Mean of Rheumatoid Arthritis Related Inpatient Visits During 12 Months Post-index Date
Description: Inpatient visits refers when participants visited hospital for formal admission. In this outcome measure, mean of number of inpatient visits related to RA during 12 months post-index were evaluated.
Time Frame: During 12 months post-index date
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Inpatient visits
Arm/Group | Tofacitinib Low OOP Cost | Tofacitinib High OOP Cost | Switch From Adalimumab to Etanercept | Switch From Adalimumab to Tofacitinib | Switch From Etanercept to Adalimumab | Switch From Etanercept to Tofacitinib
Number analyzed (Participants) | 310 | 299 | 79 | 287 | 112 | 262
Inpatient visits | 0.14 (0.42) | 0.10 (0.36) | 0.04 (0.19) | 0.08 (0.33) | 0.11 (0.47) | 0.08 (0.34)
Statistical Analysis 1: Comparison: Tofacitinib Low OOP Cost vs Tofacitinib High OOP Cost; Test type: Superiority; p = 0.3142, t-test, 2 sided
Statistical Analysis 2: Comparison: Switch From Adalimumab to Etanercept vs Switch From Adalimumab to Tofacitinib; Test type: Superiority; p = 0.2465, t-test, 2 sided
Statistical Analysis 3: Comparison: Switch From Etanercept to Adalimumab vs Switch From Etanercept to Tofacitinib; Test type: Superiority; p = 0.5933, t-test, 2 sided
Statistical Analysis 4: Comparison: Tofacitinib Low OOP Cost vs Tofacitinib High OOP Cost; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p = 0.7815, Regression, Linear; Odds Ratio (OR) = -0.0089, 95% CI 2-sided [-0.0716 to 0.0538]
Statistical Analysis 5: Comparison: Switch From Adalimumab to Etanercept vs Switch From Adalimumab to Tofacitinib; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p = 0.4446, Regression, Linear; Odds Ratio (OR) = 0.0337, 95% CI 2-sided [-0.0528 to 0.1202]
Statistical Analysis 6: Comparison: Switch From Etanercept to Adalimumab vs Switch From Etanercept to Tofacitinib; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p = 0.4733, Regression, Linear; Odds Ratio (OR) = -0.0333, 95% CI 2-sided [-0.1243 to 0.0577]

28. Secondary Outcome: Mean of Rheumatoid Arthritis Related Emergency Department (ED) Visits During 12 Months Post-index Date
Description: In this outcome measure, mean of number of emergency department visits related to RA during 12 months post-index were evaluated.
Time Frame: During 12 months post-index date
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Emergency department visits
Arm/Group | Tofacitinib Low OOP Cost | Tofacitinib High OOP Cost | Switch From Adalimumab to Etanercept | Switch From Adalimumab to Tofacitinib | Switch From Etanercept to Adalimumab | Switch From Etanercept to Tofacitinib
Number analyzed (Participants) | 310 | 299 | 79 | 287 | 112 | 262
Emergency department visits | 0.18 (0.48) | 0.12 (0.41) | 0.11 (0.39) | 0.08 (0.31) | 0.29 (1.75) | 0.23 (0.61)
Statistical Analysis 1: Comparison: Tofacitinib Low OOP Cost vs Tofacitinib High OOP Cost; Test type: Superiority; p = 0.0658, t-test, 2 sided
Statistical Analysis 2: Comparison: Switch From Adalimumab to Etanercept vs Switch From Adalimumab to Tofacitinib; Test type: Superiority; p = 0.3785, t-test, 2 sided
Statistical Analysis 3: Comparison: Switch From Etanercept to Adalimumab vs Switch From Etanercept to Tofacitinib; Test type: Superiority; p = 0.6202, t-test, 2 sided
Statistical Analysis 4: Comparison: Tofacitinib Low OOP Cost vs Tofacitinib High OOP Cost; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p = 0.2523, Regression, Linear; Odds Ratio (OR) = -0.0425, 95% CI 2-sided [-0.1154 to 0.0303]
Statistical Analysis 5: Comparison: Switch From Adalimumab to Etanercept vs Switch From Adalimumab to Tofacitinib; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p = 0.4068, Regression, Linear; Odds Ratio (OR) = -0.0388, 95% CI 2-sided [-0.1305 to 0.0529]
Statistical Analysis 6: Comparison: Switch From Etanercept to Adalimumab vs Switch From Etanercept to Tofacitinib; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p = 0.5858, Regression, Linear; Odds Ratio (OR) = 0.0706, 95% CI 2-sided [-0.1833 to 0.3244]

29. Secondary Outcome: Mean of Rheumatoid Arthritis Related Outpatient Visits During 12 Months Post-index Date
Description: Outpatient visits refers when participants visited hospital but not for formal admission. In this outcome measure, mean of number of outpatient visits related to RA during 12 months post-index were evaluated.
Time Frame: During 12 months post-index date
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Outpatient visits
Arm/Group | Tofacitinib Low OOP Cost | Tofacitinib High OOP Cost | Switch From Adalimumab to Etanercept | Switch From Adalimumab to Tofacitinib | Switch From Etanercept to Adalimumab | Switch From Etanercept to Tofacitinib
Number analyzed (Participants) | 310 | 299 | 79 | 287 | 112 | 262
Outpatient visits | 8.60 (7.17) | 8.14 (5.72) | 7.51 (5.53) | 8.06 (6.08) | 8.52 (6.68) | 8.88 (6.32)
Statistical Analysis 1: Comparison: Tofacitinib Low OOP Cost vs Tofacitinib High OOP Cost; Test type: Superiority; p = 0.3832, t-test, 2 sided
Statistical Analysis 2: Comparison: Switch From Adalimumab to Etanercept vs Switch From Adalimumab to Tofacitinib; Test type: Superiority; p = 0.4631, t-test, 2 sided
Statistical Analysis 3: Comparison: Switch From Etanercept to Adalimumab vs Switch From Etanercept to Tofacitinib; Test type: Superiority; p = 0.6202, t-test, 2 sided
Statistical Analysis 4: Comparison: Tofacitinib Low OOP Cost vs Tofacitinib High OOP Cost; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p = 0.3158, Regression, Linear; Odds Ratio (OR) = -0.5353, 95% CI 2-sided [-1.5812 to 0.5107]
Statistical Analysis 5: Comparison: Switch From Adalimumab to Etanercept vs Switch From Adalimumab to Tofacitinib; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p = 0.1016, Regression, Linear; Odds Ratio (OR) = 1.3543, 95% CI 2-sided [-0.2669 to 2.9755]
Statistical Analysis 6: Comparison: Switch From Etanercept to Adalimumab vs Switch From Etanercept to Tofacitinib; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p = 0.2576, Regression, Linear; Odds Ratio (OR) = 0.8677, 95% CI 2-sided [-0.6347 to 2.3700]

30. Secondary Outcome: Mean of Rheumatoid Arthritis Related Pharmacy Visits During 12 Months Post-index Date
Description: In this outcome measure, mean of number of pharmacy visits related to RA during 12 months post-index were evaluated.
Time Frame: During 12 months post-index date
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Pharmacy visits
Arm/Group | Tofacitinib Low OOP Cost | Tofacitinib High OOP Cost | Switch From Adalimumab to Etanercept | Switch From Adalimumab to Tofacitinib | Switch From Etanercept to Adalimumab | Switch From Etanercept to Tofacitinib
Number analyzed (Participants) | 310 | 299 | 79 | 287 | 112 | 262
Pharmacy visits | 18.76 (10.77) | 17.86 (11.08) | 19.80 (11.74) | 18.57 (10.57) | 20.13 (11.15) | 19.08 (10.59)
Statistical Analysis 1: Comparison: Tofacitinib Low OOP Cost vs Tofacitinib High OOP Cost; Test type: Superiority; p = 0.3107, t-test, 2 sided
Statistical Analysis 2: Comparison: Switch From Adalimumab to Etanercept vs Switch From Adalimumab to Tofacitinib; Test type: Superiority; p = 0.3735, t-test, 2 sided
Statistical Analysis 3: Comparison: Switch From Etanercept to Adalimumab vs Switch From Etanercept to Tofacitinib; Test type: Superiority; p = 0.3863, t-test, 2 sided
Statistical Analysis 4: Comparison: Tofacitinib Low OOP Cost vs Tofacitinib High OOP Cost; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p = 0.1918, Regression, Linear; Odds Ratio (OR) = -1.0337, 95% CI 2-sided [-2.5858 to 0.5184]
Statistical Analysis 5: Comparison: Switch From Adalimumab to Etanercept vs Switch From Adalimumab to Tofacitinib; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p = 0.4281, Regression, Linear; Odds Ratio (OR) = -0.9749, 95% CI 2-sided [-3.3864 to 1.4366]
Statistical Analysis 6: Comparison: Switch From Etanercept to Adalimumab vs Switch From Etanercept to Tofacitinib; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p = 0.1014, Regression, Linear; Odds Ratio (OR) = -1.8599, 95% CI 2-sided [-4.0854 to 0.3657]

31. Secondary Outcome: Mean of All Cause Inpatient Visits During 12 Months Pre-Index Date
Description: Inpatient visits refers when participants visited hospital for formal admission. In this outcome measure, mean of number of inpatient visits regardless of reason (including related to RA) during 12 months pre-index were evaluated.
Time Frame: During 12 months pre-index date
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Inpatient visits
Arm/Group | Tofacitinib Low OOP Cost | Tofacitinib High OOP Cost | Switch From Adalimumab to Etanercept | Switch From Adalimumab to Tofacitinib | Switch From Etanercept to Adalimumab | Switch From Etanercept to Tofacitinib
Number analyzed (Participants) | 310 | 299 | 79 | 287 | 112 | 262
Inpatient visits | 0.14 (0.39) | 0.17 (0.54) | 0.13 (0.43) | 0.15 (0.43) | 0.10 (0.46) | 0.16 (0.48)
Statistical Analysis 1: Comparison: Tofacitinib Low OOP Cost vs Tofacitinib High OOP Cost; Test type: Superiority; p = 0.4555, t-test, 2 sided
Statistical Analysis 2: Comparison: Switch From Adalimumab to Etanercept vs Switch From Adalimumab to Tofacitinib; Test type: Superiority; p = 0.7164, t-test, 2 sided
Statistical Analysis 3: Comparison: Switch From Etanercept to Adalimumab vs Switch From Etanercept to Tofacitinib; Test type: Superiority; p = 0.2456, t-test, 2 sided
Statistical Analysis 4: Comparison: Tofacitinib Low OOP Cost vs Tofacitinib High OOP Cost; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p = 0.0962, Regression, Linear; Odds Ratio (OR) = 0.0568, 95% CI 2-sided [-0.0101 to 0.1238]
Statistical Analysis 5: Comparison: Switch From Adalimumab to Etanercept vs Switch From Adalimumab to Tofacitinib; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p = 0.3844, Regression, Linear; Odds Ratio (OR) = -0.0432, 95% CI 2-sided [-0.1405 to 0.0541]
Statistical Analysis 6: Comparison: Switch From Etanercept to Adalimumab vs Switch From Etanercept to Tofacitinib; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p = 0.5899, Regression, Linear; Odds Ratio (OR) = 0.0233, 95% CI 2-sided [-0.0615 to 0.1082]

32. Secondary Outcome: Mean of All Cause Emergency Department (ED) Visits During 12 Months Pre-index Date
Description: In this outcome measure, mean of number of emergency department visits regardless of reason (including related to RA) during 12 months pre-index were evaluated.
Time Frame: During 12 months pre-index date
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Emergency department visits
Arm/Group | Tofacitinib Low OOP Cost | Tofacitinib High OOP Cost | Switch From Adalimumab to Etanercept | Switch From Adalimumab to Tofacitinib | Switch From Etanercept to Adalimumab | Switch From Etanercept to Tofacitinib
Number analyzed (Participants) | 310 | 299 | 79 | 287 | 112 | 262
Emergency department visits | 0.55 (0.95) | 0.47 (1.34) | 0.52 (1.27) | 0.47 (1.09) | 0.63 (2.76) | 0.60 (1.46)
Statistical Analysis 1: Comparison: Tofacitinib Low OOP Cost vs Tofacitinib High OOP Cost; Test type: Superiority; p = 0.4133, t-test, 2 sided
Statistical Analysis 2: Comparison: Switch From Adalimumab to Etanercept vs Switch From Adalimumab to Tofacitinib; Test type: Superiority; p = 0.7171, t-test, 2 sided
Statistical Analysis 3: Comparison: Switch From Etanercept to Adalimumab vs Switch From Etanercept to Tofacitinib; Test type: Superiority; p = 0.8609, t-test, 2 sided
Statistical Analysis 4: Comparison: Tofacitinib Low OOP Cost vs Tofacitinib High OOP Cost; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p = 0.6224, Regression, Linear; Odds Ratio (OR) = -0.0445, 95% CI 2-sided [-0.2218 to 0.1327]
Statistical Analysis 5: Comparison: Switch From Adalimumab to Etanercept vs Switch From Adalimumab to Tofacitinib; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p = 0.5655, Regression, Linear; Odds Ratio (OR) = -0.0884, 95% CI 2-sided [-0.3900 to 0.2132]
Statistical Analysis 6: Comparison: Switch From Etanercept to Adalimumab vs Switch From Etanercept to Tofacitinib; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p = 0.4044, Regression, Linear; Odds Ratio (OR) = 0.1809, 95% CI 2-sided [-0.2444 to 0.6062]

33. Secondary Outcome: Mean of All Cause Outpatient Visits During 12 Months Pre-Index Date
Description: Outpatient visits refers when participants visited hospital but not for formal admission. In this outcome measure, mean of number of outpatient visits regardless of reason (including related to RA) during 12 months pre-index were evaluated.
Time Frame: During 12 months pre-index date
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Outpatient visits
Arm/Group | Tofacitinib Low OOP Cost | Tofacitinib High OOP Cost | Switch From Adalimumab to Etanercept | Switch From Adalimumab to Tofacitinib | Switch From Etanercept to Adalimumab | Switch From Etanercept to Tofacitinib
Number analyzed (Participants) | 310 | 299 | 79 | 287 | 112 | 262
Outpatient visits | 31.70 (22.60) | 27.26 (19.81) | 28.48 (23.30) | 29.92 (20.62) | 27.23 (18.21) | 31.45 (22.50)
Statistical Analysis 1: Comparison: Tofacitinib Low OOP Cost vs Tofacitinib High OOP Cost; Test type: Superiority; p = 0.0104, t-test, 2 sided
Statistical Analysis 2: Comparison: Switch From Adalimumab to Etanercept vs Switch From Adalimumab to Tofacitinib; Test type: Superiority; p = 0.5949, t-test, 2 sided
Statistical Analysis 3: Comparison: Switch From Etanercept to Adalimumab vs Switch From Etanercept to Tofacitinib; Test type: Superiority; p = 0.0801, t-test, 2 sided
Statistical Analysis 4: Comparison: Tofacitinib Low OOP Cost vs Tofacitinib High OOP Cost; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p = 0.0072, Regression, Linear; Odds Ratio (OR) = -3.7075, 95% CI 2-sided [-6.4110 to -1.0040]
Statistical Analysis 5: Comparison: Switch From Adalimumab to Etanercept vs Switch From Adalimumab to Tofacitinib; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p = 0.5406, Regression, Linear; Odds Ratio (OR) = -1.4296, 95% CI 2-sided [-6.0080 to 3.1489]
Statistical Analysis 6: Comparison: Switch From Etanercept to Adalimumab vs Switch From Etanercept to Tofacitinib; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p = 0.8603, Regression, Linear; Odds Ratio (OR) = -0.3527, 95% CI 2-sided [-4.2790 to 3.5737]

34. Secondary Outcome: Mean of All Cause Pharmacy Visits During 12 Months Pre-index Date
Description: In this outcome measure, mean of number of pharmacy visits regardless of reason (including related to RA) during 12 months pre-index were evaluated.
Time Frame: During 12 months pre-index date
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Pharmacy visits
Arm/Group | Tofacitinib Low OOP Cost | Tofacitinib High OOP Cost | Switch From Adalimumab to Etanercept | Switch From Adalimumab to Tofacitinib | Switch From Etanercept to Adalimumab | Switch From Etanercept to Tofacitinib
Number analyzed (Participants) | 310 | 299 | 79 | 287 | 112 | 262
Pharmacy visits | 41.69 (30.60) | 40.56 (27.62) | 42.47 (27.03) | 46.24 (29.26) | 41.83 (28.58) | 47.29 (33.67)
Statistical Analysis 1: Comparison: Tofacitinib Low OOP Cost vs Tofacitinib High OOP Cost; Test type: Superiority; p = 0.6344, t-test, 2 sided
Statistical Analysis 2: Comparison: Switch From Adalimumab to Etanercept vs Switch From Adalimumab to Tofacitinib; Test type: Superiority; p = 0.3037, t-test, 2 sided
Statistical Analysis 3: Comparison: Switch From Etanercept to Adalimumab vs Switch From Etanercept to Tofacitinib; Test type: Superiority; p = 0.1344, t-test, 2 sided
Statistical Analysis 4: Comparison: Tofacitinib Low OOP Cost vs Tofacitinib High OOP Cost; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p = 0.5092, Regression, Linear; Odds Ratio (OR) = 1.2586, 95% CI 2-sided [-2.4787 to 4.9958]
Statistical Analysis 5: Comparison: Switch From Adalimumab to Etanercept vs Switch From Adalimumab to Tofacitinib; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p = 0.8047, Regression, Linear; Odds Ratio (OR) = -0.7696, 95% CI 2-sided [-6.8683 to 5.3292]
Statistical Analysis 6: Comparison: Switch From Etanercept to Adalimumab vs Switch From Etanercept to Tofacitinib; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p = 0.9757, Regression, Linear; Odds Ratio (OR) = 0.0940, 95% CI 2-sided [-5.9628 to 6.1507]

35. Secondary Outcome: Mean of All Cause Inpatient Visits During 12 Months Post-index Date
Description: Inpatient visits refers when participants visited hospital for formal admission. In this outcome measure, mean of number of inpatient visits regardless of reason (including related to RA) during 12 months post-index were evaluated.
Time Frame: During 12 months post-index date
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Inpatient visits
Arm/Group | Tofacitinib Low OOP Cost | Tofacitinib High OOP Cost | Switch From Adalimumab to Etanercept | Switch From Adalimumab to Tofacitinib | Switch From Etanercept to Adalimumab | Switch From Etanercept to Tofacitinib
Number analyzed (Participants) | 310 | 299 | 79 | 287 | 112 | 262
Inpatient visits | 0.24 (0.58) | 0.16 (0.53) | 0.14 (0.71) | 0.14 (0.48) | 0.24 (1.21) | 0.25 (0.87)
Statistical Analysis 1: Comparison: Tofacitinib Low OOP Cost vs Tofacitinib High OOP Cost; Test type: Superiority; p = 0.0839, t-test, 2 sided
Statistical Analysis 2: Comparison: Switch From Adalimumab to Etanercept vs Switch From Adalimumab to Tofacitinib; Test type: Superiority; p = 0.9577, t-test, 2 sided
Statistical Analysis 3: Comparison: Switch From Etanercept to Adalimumab vs Switch From Etanercept to Tofacitinib; Test type: Superiority; p = 0.9497, t-test, 2 sided
Statistical Analysis 4: Comparison: Tofacitinib Low OOP Cost vs Tofacitinib High OOP Cost; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p = 0.4873, Regression, Linear; Odds Ratio (OR) = -0.0310, 95% CI 2-sided [-0.1185 to 0.0565]
Statistical Analysis 5: Comparison: Switch From Adalimumab to Etanercept vs Switch From Adalimumab to Tofacitinib; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p = 0.6780, Regression, Linear; Odds Ratio (OR) = -0.0312, 95% CI 2-sided [-0.1783 to 0.1159]
Statistical Analysis 6: Comparison: Switch From Etanercept to Adalimumab vs Switch From Etanercept to Tofacitinib; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p = 0.9327, Regression, Linear; Odds Ratio (OR) = 0.0099, 95% CI 2-sided [-0.2207 to 0.2406]

36. Secondary Outcome: Mean of All Cause Emergency Department (ED) Visits During 12 Months Post-index Date
Description: In this outcome measure, mean of number of emergency department visits regardless of reason (including related to RA) during 12 months post-index were evaluated.
Time Frame: During 12 months post-index date
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Emergency department visits
Arm/Group | Tofacitinib Low OOP Cost | Tofacitinib High OOP Cost | Switch From Adalimumab to Etanercept | Switch From Adalimumab to Tofacitinib | Switch From Etanercept to Adalimumab | Switch From Etanercept to Tofacitinib
Number analyzed (Participants) | 310 | 299 | 79 | 287 | 112 | 262
Emergency department visits | 0.68 (1.25) | 0.41 (0.89) | 0.52 (0.96) | 0.44 (1.04) | 1.04 (7.23) | 0.81 (1.63)
Statistical Analysis 1: Comparison: Tofacitinib Low OOP Cost vs Tofacitinib High OOP Cost; Test type: Superiority; p = 0.0021, t-test, 2 sided
Statistical Analysis 2: Comparison: Switch From Adalimumab to Etanercept vs Switch From Adalimumab to Tofacitinib; Test type: Superiority; p = 0.5396, t-test, 2 sided
Statistical Analysis 3: Comparison: Switch From Etanercept to Adalimumab vs Switch From Etanercept to Tofacitinib; Test type: Superiority; p = 0.6121, t-test, 2 sided
Statistical Analysis 4: Comparison: Tofacitinib Low OOP Cost vs Tofacitinib High OOP Cost; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p = 0.0303, Regression, Linear; Odds Ratio (OR) = -0.1895, 95% CI 2-sided [-0.3610 to -0.0181]
Statistical Analysis 5: Comparison: Switch From Adalimumab to Etanercept vs Switch From Adalimumab to Tofacitinib; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p = 0.1807, Regression, Linear; Odds Ratio (OR) = -0.1901, 95% CI 2-sided [-0.4685 to 0.0883]
Statistical Analysis 6: Comparison: Switch From Etanercept to Adalimumab vs Switch From Etanercept to Tofacitinib; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p = 0.7445, Regression, Linear; Odds Ratio (OR) = 0.1594, 95% CI 2-sided [-0.7991 to 1.1178]

37. Secondary Outcome: Mean of All Cause Outpatient Visits During 12 Months Post-index Date
Description: Outpatient visits refers when participants visited hospital but not for formal admission. In this outcome measure, mean of number of outpatient visits regardless of reason (including related to RA) during 12 months post-index were evaluated.
Time Frame: During 12 months post-index date
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Outpatient visits
Arm/Group | Tofacitinib Low OOP Cost | Tofacitinib High OOP Cost | Switch From Adalimumab to Etanercept | Switch From Adalimumab to Tofacitinib | Switch From Etanercept to Adalimumab | Switch From Etanercept to Tofacitinib
Number analyzed (Participants) | 310 | 299 | 79 | 287 | 112 | 262
Outpatient visits | 33.30 (29.56) | 27.16 (21.30) | 27.00 (21.04) | 28.89 (22.48) | 28.39 (22.90) | 32.76 (27.14)
Statistical Analysis 1: Comparison: Tofacitinib Low OOP Cost vs Tofacitinib High OOP Cost; Test type: Superiority; p = 0.0035, t-test, 2 sided
Statistical Analysis 2: Comparison: Switch From Adalimumab to Etanercept vs Switch From Adalimumab to Tofacitinib; Test type: Superiority; p = 0.5040, t-test, 2 sided
Statistical Analysis 3: Comparison: Switch From Etanercept to Adalimumab vs Switch From Etanercept to Tofacitinib; Test type: Superiority; p = 0.1366, t-test, 2 sided
Statistical Analysis 4: Comparison: Tofacitinib Low OOP Cost vs Tofacitinib High OOP Cost; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p = 0.0820, Regression, Linear; Odds Ratio (OR) = -3.4084, 95% CI 2-sided [-7.2497 to 0.4330]
Statistical Analysis 5: Comparison: Switch From Adalimumab to Etanercept vs Switch From Adalimumab to Tofacitinib; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p = 0.5845, Regression, Linear; Odds Ratio (OR) = -1.5342, 95% CI 2-sided [-7.0336 to 3.9652]
Statistical Analysis 6: Comparison: Switch From Etanercept to Adalimumab vs Switch From Etanercept to Tofacitinib; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p = 0.7284, Regression, Linear; Odds Ratio (OR) = 0.9870, 95% CI 2-sided [-4.5830 to 6.5570]

38. Secondary Outcome: Mean of All Cause Pharmacy Visits During 12 Months Post-index Date
Description: In this outcome measure, mean of number of pharmacy visits regardless of reason (including related to RA) during 12 months post-index were evaluated.
Time Frame: During 12 months post-index date
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Pharmacy visits
Arm/Group | Tofacitinib Low OOP Cost | Tofacitinib High OOP Cost | Switch From Adalimumab to Etanercept | Switch From Adalimumab to Tofacitinib | Switch From Etanercept to Adalimumab | Switch From Etanercept to Tofacitinib
Number analyzed (Participants) | 310 | 299 | 79 | 287 | 112 | 262
Pharmacy visits | 49.32 (34.05) | 45.25 (28.85) | 46.33 (27.41) | 47.70 (30.26) | 45.70 (27.46) | 50.09 (31.99)
Statistical Analysis 1: Comparison: Tofacitinib Low OOP Cost vs Tofacitinib High OOP Cost; Test type: Superiority; p = 0.1125, t-test, 2 sided
Statistical Analysis 2: Comparison: Switch From Adalimumab to Etanercept vs Switch From Adalimumab to Tofacitinib; Test type: Superiority; p = 0.7156, t-test, 2 sided
Statistical Analysis 3: Comparison: Switch From Etanercept to Adalimumab vs Switch From Etanercept to Tofacitinib; Test type: Superiority; p = 0.2056, t-test, 2 sided
Statistical Analysis 4: Comparison: Tofacitinib Low OOP Cost vs Tofacitinib High OOP Cost; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p = 0.4288, Regression, Linear; Odds Ratio (OR) = -1.8061, 95% CI 2-sided [-6.2797 to 2.6675]
Statistical Analysis 5: Comparison: Switch From Adalimumab to Etanercept vs Switch From Adalimumab to Tofacitinib; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p = 0.6303, Regression, Linear; Odds Ratio (OR) = -1.6946, 95% CI 2-sided [-8.5962 to 5.2069]
Statistical Analysis 6: Comparison: Switch From Etanercept to Adalimumab vs Switch From Etanercept to Tofacitinib; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p = 0.7477, Regression, Linear; Odds Ratio (OR) = -0.9873, 95% CI 2-sided [-7.0028 to 5.0281]

39. Secondary Outcome: Mean of Rheumatoid Arthritis Related Total Health Care Cost During 12 Months Pre-index Date
Description: Total health care cost related to RA was calculated as sum of medical (outpatient, inpatient and emergency visit) cost and treatment costs (pharmacy cost) related to rheumatoid arthritis.
Time Frame: During 12 months pre-index date
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Dollars
Arm/Group | Tofacitinib Low OOP Cost | Tofacitinib High OOP Cost | Switch From Adalimumab to Etanercept | Switch From Adalimumab to Tofacitinib | Switch From Etanercept to Adalimumab | Switch From Etanercept to Tofacitinib
Number analyzed (Participants) | 310 | 299 | 79 | 287 | 112 | 262
Dollars | 6316.86 (14673.52) | 7414.19 (16892.85) | 16343.48 (15762.03) | 27375.50 (20613.83) | 18432.35 (15754.60) | 22777.88 (16633.19)
Statistical Analysis 1: Comparison: Tofacitinib Low OOP Cost vs Tofacitinib High OOP Cost; Test type: Superiority; p = 0.3919, t-test, 2 sided
Statistical Analysis 2: Comparison: Switch From Adalimumab to Etanercept vs Switch From Adalimumab to Tofacitinib; Test type: Superiority; p < 0.0001, t-test, 2 sided
Statistical Analysis 3: Comparison: Switch From Etanercept to Adalimumab vs Switch From Etanercept to Tofacitinib; Test type: Superiority; p = 0.0193, t-test, 2 sided
Statistical Analysis 4: Comparison: Tofacitinib Low OOP Cost vs Tofacitinib High OOP Cost; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p = 0.0570, Regression, Linear; Cost Ratio = 1.2232, 95% CI 2-sided [0.9940 to 1.5053] — Since health care costs were skewed, hence estimated cost was modeled using a generalized linear model (GLM). Coefficients from a generalized linear model were estimated as cost ratios
Statistical Analysis 5: Comparison: Switch From Adalimumab to Etanercept vs Switch From Adalimumab to Tofacitinib; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p < 0.0001, Regression, Linear; Cost Ratio = 1.8479, 95% CI 2-sided [1.4378 to 2.3749] — Since health care costs were skewed, hence estimated cost was modeled using a GLM. Coefficients from a generalized linear model were estimated as cost ratios
Statistical Analysis 6: Comparison: Switch From Etanercept to Adalimumab vs Switch From Etanercept to Tofacitinib; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p = 0.0924, Regression, Linear; Cost Ratio = 1.1868, 95% CI 2-sided [0.9722 to 1.4487] — [estimate comment as in outcome 39, analysis 5]

40. Secondary Outcome: Mean of Rheumatoid Arthritis Related Total Health Care Cost During 12 Months Post-index Date
Description: as for outcome 39
Time Frame: During 12 months post-index date
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Dollars
Arm/Group | Tofacitinib Low OOP Cost | Tofacitinib High OOP Cost | Switch From Adalimumab to Etanercept | Switch From Adalimumab to Tofacitinib | Switch From Etanercept to Adalimumab | Switch From Etanercept to Tofacitinib
Number analyzed (Participants) | 310 | 299 | 79 | 287 | 112 | 262
Dollars | 35601.32 (22826.82) | 34503.47 (31045.94) | 34010.25 (17628.32) | 37431.71 (21525.40) | 40027.03 (20886.32) | 36963.17 (18806.38)
Statistical Analysis 1: Comparison: Tofacitinib Low OOP Cost vs Tofacitinib High OOP Cost; Test type: Superiority; p = 0.6184, t-test, 2 sided
Statistical Analysis 2: Comparison: Switch From Adalimumab to Etanercept vs Switch From Adalimumab to Tofacitinib; Test type: Superiority; p = 0.1952, t-test, 2 sided
Statistical Analysis 3: Comparison: Switch From Etanercept to Adalimumab vs Switch From Etanercept to Tofacitinib; Test type: Superiority; p = 0.1638, t-test, 2 sided
Statistical Analysis 4: Comparison: Tofacitinib Low OOP Cost vs Tofacitinib High OOP Cost; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p = 0.6732, Regression, Linear; Cost Ratio = 0.9773, 95% CI 2-sided [0.8782 to 1.0875] — [estimate comment as in outcome 39, analysis 5]
Statistical Analysis 5: Comparison: Switch From Adalimumab to Etanercept vs Switch From Adalimumab to Tofacitinib; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p = 0.6345, Regression, Linear; Cost Ratio = 0.9629, 95% CI 2-sided [0.8240 to 1.1253] — [estimate comment as in outcome 39, analysis 5]
Statistical Analysis 6: Comparison: Switch From Etanercept to Adalimumab vs Switch From Etanercept to Tofacitinib; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p = 0.0029, Regression, Linear; Cost Ratio = 0.8327, 95% CI 2-sided [0.7380 to 0.9395] — [estimate comment as in outcome 39, analysis 5]

41. Secondary Outcome: All Cause Total Health Care Cost During 12 Months Pre-index Date
Description: All cause total health care cost was calculated as sum of medical (outpatient, inpatient and emergency visit) cost and treatment cost (pharmacy cost) regardless of reason including RA.
Time Frame: During 12 months pre-index date
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Dollars
Arm/Group | Tofacitinib Low OOP Cost | Tofacitinib High OOP Cost | Switch From Adalimumab to Etanercept | Switch From Adalimumab to Tofacitinib | Switch From Etanercept to Adalimumab | Switch From Etanercept to Tofacitinib
Number analyzed (Participants) | 310 | 299 | 79 | 287 | 112 | 262
Dollars | 22626.74 (43882.45) | 19514.09 (29958.63) | 25944.31 (21338.45) | 38749.72 (28956.92) | 29643.91 (31487.43) | 36152.42 (30954.57)
Statistical Analysis 1: Comparison: Tofacitinib Low OOP Cost vs Tofacitinib High OOP Cost; Test type: Superiority; p = 0.3087, t-test, 2 sided
Statistical Analysis 2: Comparison: Switch From Adalimumab to Etanercept vs Switch From Adalimumab to Tofacitinib; Test type: Superiority; p = 0.0003, t-test, 2 sided
Statistical Analysis 3: Comparison: Switch From Etanercept to Adalimumab vs Switch From Etanercept to Tofacitinib; Test type: Superiority; p = 0.0647, t-test, 2 sided
Statistical Analysis 4: Comparison: Tofacitinib Low OOP Cost vs Tofacitinib High OOP Cost; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p = 0.7684, Regression, Linear; Cost Ratio = 0.9762, 95% CI 2-sided [0.8316 to 1.1460] — [estimate comment as in outcome 39, analysis 5]
Statistical Analysis 5: Comparison: Switch From Adalimumab to Etanercept vs Switch From Adalimumab to Tofacitinib; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p = 0.0012, Regression, Linear; Cost Ratio = 1.3862, 95% CI 2-sided [1.1379 to 1.6886] — [estimate comment as in outcome 39, analysis 5]
Statistical Analysis 6: Comparison: Switch From Etanercept to Adalimumab vs Switch From Etanercept to Tofacitinib; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p = 0.9422, Regression, Linear; Cost Ratio = 1.0065, 95% CI 2-sided [0.8452 to 1.1985] — [estimate comment as in outcome 39, analysis 5]

42. Secondary Outcome: All Cause Total Health Care Cost During 12 Months Post-index Date
Description: as for outcome 41
Time Frame: During 12 months post-index date
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Dollars
Arm/Group | Tofacitinib Low OOP Cost | Tofacitinib High OOP Cost | Switch From Adalimumab to Etanercept | Switch From Adalimumab to Tofacitinib | Switch From Etanercept to Adalimumab | Switch From Etanercept to Tofacitinib
Number analyzed (Participants) | 310 | 299 | 79 | 287 | 112 | 262
Dollars | 56515.65 (78961.26) | 46126.57 (39998.62) | 50343.02 (68582.27) | 49109.94 (29561.43) | 56302.76 (61613.45) | 56786.41 (57000.99)
Statistical Analysis 1: Comparison: Tofacitinib Low OOP Cost vs Tofacitinib High OOP Cost; Test type: Superiority; p = 0.0421, t-test, 2 sided
Statistical Analysis 2: Comparison: Switch From Adalimumab to Etanercept vs Switch From Adalimumab to Tofacitinib; Test type: Superiority; p = 0.8137, t-test, 2 sided
Statistical Analysis 3: Comparison: Switch From Etanercept to Adalimumab vs Switch From Etanercept to Tofacitinib; Test type: Superiority; p = 0.9416, t-test, 2 sided
Statistical Analysis 4: Comparison: Tofacitinib Low OOP Cost vs Tofacitinib High OOP Cost; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p = 0.3190, Regression, Linear; Cost Ratio = 0.9515, 95% CI 2-sided [0.8628 to 1.0493] — [estimate comment as in outcome 39, analysis 5]
Statistical Analysis 5: Comparison: Switch From Adalimumab to Etanercept vs Switch From Adalimumab to Tofacitinib; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p = 0.1368, Regression, Linear; Cost Ratio = 0.8991, 95% CI 2-sided [0.7815 to 1.0343] — [estimate comment as in outcome 39, analysis 5]
Statistical Analysis 6: Comparison: Switch From Etanercept to Adalimumab vs Switch From Etanercept to Tofacitinib; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p = 0.0231, Regression, Linear; Cost Ratio = 0.8514, 95% CI 2-sided [0.7411 to 0.9782] — [estimate comment as in outcome 39, analysis 5]

ADVERSE EVENTS:
Time Frame: Not applicable as safety data was not planned to be collected and evaluated during the study
Description: Study used de-identified structured data. Minimum criteria for reporting an adverse event (identifiable participant, identifiable reporter, a suspect product/treatment, and event) could not be met. Hence, due to the nature of claims database from which data were queried, no adverse events were collected.
Arm/Group | Tofacitinib Low OOP Cost | Tofacitinib High OOP Cost | Switch From Adalimumab to Etanercept | Switch From Adalimumab to Tofacitinib | Switch From Etanercept to Adalimumab | Switch From Etanercept to Tofacitinib
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Prioritization for outcome measures was per study team's discretion.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-07): https://cdn.clinicaltrials.gov/large-docs/21/NCT04047121/Prot_SAP_000.pdf